#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for 201789: A Phase 1/2, Double-Blind, Placebo-Controlled Study of the Pharmacokinetics, Safety and Tolerability of GSK3196165 in Combination with Methotrexate Therapy, in Japanese Subjects with Active Moderate-Severe Rheumatoid Arthritis Despite Treatment with Methotrexate. |
|---|---|---|
| <b>Compound Number</b> | : | GSK3196165 |
| <b>Effective Date</b> | : | 24-JAN-2018 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 201789.
- This RAP is intended to describe the pharmacokinetic, safety, immunogenicity, efficacy, pharmacodynamic and pharmacokinetic/pharmacodynamic analyses required for the study.
- This version includes amendments to the originally approved RAP.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Approver | Date | Approval<br>Method |
|---|---|---|
| PPD | | |
| Biostatistics Group2, Biomedical Data Sciences, | | |
| Japan | | |
| PPD | | |
| Manager, Clinical Pharmacology & Science | 17-Jan-2018 | Email |
| Promotion Office, Medicines Development | | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### The GlaxoSmithKline group of companies

### **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Immuno-Inflammation, Dermatology TA Office, | 18-Jan-2018 | Email |
| Medicines Development, Japan | | |
| Clinical Operations Dept., Japan | 19-Jan-2018 | Email |
| Data Practice Group, Biomedical Data Sciences<br>Dept., Japan | 19-Jan-2018 | Email |
| Medical Writing Office, Medicines Development, Japan | 19-Jan-2018 | Email |
| Clinical Pharmacology & Science Promotion Office, Medicines Development, Japan | 19-Jan-2018 | Email |
| Statistical Programming & Reporting Group, Biomedical Data Sciences, Japan | 19-Jan-2018 | Email |

### **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Manager, Biostatistics Group2, Biomedical Data Sciences, Japan | 24-Jan-2018 | Email |
| Manager, Statistical Programming & Reporting Group, Biomedical Data Sciences, Japan | 23-Jan-2018 | Email |

### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | | & ANALYSIS PLAN SYNPOSISmendments | |
| 2. | <ul><li>2.1. Chang</li><li>2.2. Study</li><li>2.3. Study</li></ul> | F KEY PROTOCOL INFORMATIONes to the Protocol Defined Statistical Analysis Plan | 8<br>8<br>9 |
| 3. | | IALYSESnalyses | |
| 4. | | OPULATIONSol Deviations | |
| 5. | | TIONS FOR DATA ANALYSES AND DATA HANDLING | 11 |
| 6. | | PLATION ANALYSES ew of Planned Analyses Demographic Characteristics Baseline Efficacy Parameters Rheumatoid Factor and Anti-cyclic Citrullinated Protein Antibody RA disease history Corticosteroid use Exposure 6.1.6.1. GSK3196165 6.1.6.2. MTX | 11<br>13<br>13<br>13<br>13<br>14 |
| 7. | 7.1. Pharm 7.1.1. | ATISTICAL ANALYSES | 14<br>14<br>15<br>15 |
| | 7.2. Safety 7.2.1. | Analyses | 17 |
| 8. | | 8.1.1.1. Pulmonary assessment | 18<br>19<br>20 |

### **CONFIDENTIAL**

| | | 0.4.0 | | 0.4 |
|---|---|---|---|---|
| | 8.2. | | Immunogenicity Analyses | |
| | 0.2. | | Analyses | |
| | | | Overview of Planned Efficacy Analyses | |
| | | | DAS28 (CRP) | |
| | | , | 8.2.2.1. Planned Efficacy Statistical Analyses | 23 |
| 9. | EXPLO | PRATORY | STATISTICAL ANALYSES | 25 |
| | 9.1. | Overview | of Planned Exploratory Analyses | 25 |
| | | 9.1.1. | ACR 20/50/70 response | 26 |
| | | 9.1.2. | DAS28 (ESR) | 26 |
| | | | SDAI, CDAI and FACIT-Fatigue | 26 |
| | | 9.1.4. | Categorical DAS28 Response | 27 |
| | | 9.1.5. | DAS28 Remission | 27 |
| | | | Other endpoints | |
| | 9.2. | | odynamic and Biomarker Analyses | 28 |
| | | | Overview of Planned Pharmacodynamic and Biomarker | 00 |
| | 0.0 | | Analyses | |
| | 9.3. | Pharmaco | okinetic / Pharmacodynamic Analyses | 28 |
| 10. | REFER | RENCES | | 30 |
| 11. | | | | |
| | 11.1. | | 1: Time & Events | |
| | | | Protocol Defined Time & Events | |
| | 11.2. | | 2: Assessment Windows | |
| | 11.3. | <b>Appendix</b> | 3: Treatment States and Phases | 38 |
| | | | 11.3.1.1. Treatment States for Concomitant Medications | |
| | | | for Rheumatoid Arthritis (CONMEDS RA) Data | 38 |
| | | | 11.3.1.2. Treatment States for AE Data | 39 |
| | 11.4. | | 4: Data Display Standards & Handling Conventions | |
| | | | Study Treatment & Sub-group Display Descriptors | |
| | | 11.4.2. | Baseline Definition & Derivations | 40 |
| | | | 11.4.2.1. Baseline Definitions | 40 |
| | | | 11.4.2.2. Derivations and Handling of Missing Baseline | |
| | | | Data | 40 |
| | | | Reporting Process & Standards | |
| | 11.5. | | 5: Derived and Transformed Data | |
| | | | General | |
| | | | Study Population | |
| | | | Safety | |
| | | | Efficacy | |
| | | | Immunogenicity | |
| | 11.6. | | 6: Premature Withdrawals & Handling of Missing Data | |
| | | | Premature Withdrawals | |
| | | | Handling of Missing Data | |
| | | | 11.6.2.1. Handling of Partial Dates | 58 |
| | | | 11.6.2.2. Handling of Missing Data for Statistical | |
| | | | Analysis | |
| | 11.7. | | 7: Multiple Comparisons & Multiplicity | 59 |
| | 11.8. | | 8: Model Checking and Diagnostics for Statistical | |
| | | Analyses. | | 60 |
| | | 11.8.1. | Statistical Analysis Assumptions | 60 |

### **CONFIDENTIAL**

| 11.9. | Appendix | ⟨ 9 – Abbreviations & Trade Marks | 61 |
|---|---|---|---|
| | 11.9.1. | Abbreviations | 61 |
| | 11.9.2. | Trademarks | 62 |
| 11.10. | Appendix | Control of Data Displays C | 63 |
| | 11.10.1. | Data Display Numbering | 63 |
| | 11.10.2. | Deliverable | 63 |
| | 11.10.3. | Study Population Tables | 64 |
| | 11.10.4. | Efficacy Tables | 66 |
| | 11.10.5. | Efficacy Figures | 69 |
| | 11.10.6. | Safety Tables | 72 |
| | 11.10.7. | Pharmacokinetic Tables | 75 |
| | 11.10.8. | Pharmacokinetic Figures | 76 |
| | 11.10.9. | Pharmacodynamic and Biomarker Tables | 77 |
| | 11.10.10 | .Pharmacodynamic and Biomarker Figures | 79 |
| | | .Pharmacokinetic / Pharmacodynamic Figures | |
| | | .ICH Listings | |
| | 11.10.13 | .Non-ICH listings | 92 |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | <ul> <li>This RAP describes all planned analyses and outputs required for the final<br/>Clinical Study Report (CSR) of study 201789.</li> </ul> |
| Protocol | This RAP is based on the protocol [(Dated: 27/SEP/2016) of study 201789 (GSK Document No. : 2016N278580_01] and eCRF. |
| Primary<br>Objective | <ul> <li>To assess the pharmacokinetics of GSK3196165 in Japanese rheumatoid arthritis (RA) subjects</li> <li>To assess the safety and tolerability of GSK3196165 in combination with methotrexate (MTX) therapy in Japanese RA subjects.</li> </ul> |
| Primary<br>Endpoint | <ul> <li>Pharmacokinetic (PK) parameters of GSK3196165 calculated from sparse sampling concentrations.</li> <li>Incidence of adverse events (AEs), serious adverse events (SAEs) and AEs of special interest.</li> </ul> |
| Study Design | This is a randomized, double-blind, parallel group, 3 dosage level, placebo-<br>controlled, Phase 1/2 study in Japanese subjects with active moderate-<br>severe RA despite treatment with MTX. |
| Planned<br>Analyses | Final analyses will be performed according to the steps described in Section 3.1. All decisions regarding final analyses, as defined in this RAP document, will be made prior to Database Freeze (unblinding) of the study data. |
| Analysis<br>Populations | <ul> <li>The Intent to Treat (ITT) population consists of all subjects who were randomized to treatment and receive at least one dose of study treatment. This population will be used for the efficacy and safety analyses.</li> <li>PK population consists of all GSK3196165-treated subjects from whom PK samples are collected and analyzed.</li> </ul> |
| Hypothesis | No formal hypotheses will be tested. |
| Primary<br>Analyses(PK) | For serum concentration of GSK3196165 over time, individual data will be listed and presented in graphical form, and summary statistics at each time point will be calculated by each dose level. The following PK variables after the last dosing will be derived by non-compartmental analysis as applicable and as data allowed: Cmax, tmax, AUCtau, AUC(0-t), AUC(0-inf), and t1/2. For PK parameters, summary statistics will be calculated by each dose level, and scatter plots against the dose level will be generated. Dose proportionality will also be assessed with the power model. |
| Primary<br>analyses(Safety<br>and Tolerability) | All AEs will be coded using MedDRA and summarized by System Organ Class (SOC) and Preferred Term (PT). The number and percentage of subjects with any AEs will be summarized by dose. The study treatment-elated AEs, SAEs, AEs leading to discontinuation of study treatment, and AEs of special interest will be reported separately. |

### 1.1. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Plan_Study2 | 201789_Final [23-MAY-2017] |
| Reporting and Analysis Plan_Study201789_final_Amend 1 [04-OCT-2017] | |
| Section 3.1 and Section 3.2 | Removed these sections because the planned interim |
| | analyses have been canceled. |
| Section 3.3 | Removed this section and added the unblinding process. |
| Section 3.1 | Removed "(interim and final)". |
| Section 8.2.1 | Added the listing of change from baseline in DAS28(CRP) |
| Section 9.1 | Added the listings of ACR response, Categorical DAS28 |
| Section 9.1 | response and DAS28 remission Added the listing of change from baseline in DAS28(ESR) |
| Section 11.4.3 | Removed the Reporting area for interim analyses |
| Section 11.4.3 | Amended the area for final reporting |
| Section 11.10.1 | Amended the Numbering according to the change of the TLF. |
| Section 11.10.2 | Removed the delivery description for interim analyses |
| Section 11.10.3, Section 11.10.4, | Removed the TOC of TLF for interim analyses. |
| Section 11.10.5, Section 11.10.6 and | Tromovou and 100 of 121 for interim unary 500. |
| Section 11.10.12 | |
| Section 11.10.9 and Section 11.10.10 | Amended the TOC to simplify it. |
| Section 11.10.11 | Amended the typos. |
| Section 11.10.12 | Added the listings of ACR20/50/70, Categorical DAS28 |
| | response and DAS28 remission |
| Reporting and Analysis Plan_Study2 | 201789_final_Amend 2 [24-Jan-2018] |
| Section 4. | Removed "valid" to avoid misunderstanding. |
| Section 6.1.3. | Added the description of RF and ACPA analyses. |
| Section 7.1.3.2. | Added one pharmacokinetic parameter "AUC(0-t)" for dose |
| | proportionality. |
| Section 7.2.1. | Added 3 AESI listings (Infection, Hypersensitivity Reactions |
| | and Injection Site Reaction) |
| Section 8.1.1. | Removed the summary of change from baseline in Borg scale |
| 0 " 010 | becase this variable is categorical. |
| Section 8.1.3. | Added the details of Immunogenicity analyses because of |
| Castian 44.0 | clarification of data in detail |
| Section 11.2. | Clarified that early withdrawal visits will be included for Assessment Windows. |
| Section 11.5.2 | Added the reference date for Age calculation |
| Section 11.5.2 | Added the definitions of Age Group and Age Category |
| Section 11.5.2 | Amended the procedure for average daily dose of OCS to |
| | calculate it at only each scheduled visit. |
| Section 11.5.3 | Amended the specification of AESI because the procedure to |
| | specify AESI was changed. |
| Section 11.5.4 | Clarified that when calculating ACR, Patient's Assessment for |
| | Arthritis Pain "at this time" will be used. |
| Section 11.5.4 | Amended the typos in SJC and TJC section. |
| Section 11.10. | Amended Shell IDs and titles. |
| | Added some displays. |

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol [(Dated: 27/SEP/2016)].

### 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the PK of GSK3196165 in<br>Japanese RA subjects | PK parameters of GSK3196165 calculated from sparse sampling concentrations |
| To assess the safety and tolerability of<br>GSK 3196165 in combination with<br>MTX therapy in Japanese RA subjects | Incidence of AEs, SAEs and AEs of special interest |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To assess the safety other than primary endpoints</li> <li>To assess the efficacy in Japanese RA subjects</li> </ul> | <ul> <li>Vital signs, 12-lead ECG and laboratory assessment</li> <li>Immunogenicity (anti-GSK3196165 antibody)</li> <li>Change from baseline in Disease Activity Score 28 [DAS28(CRP)] at all assessment timepoints</li> </ul> |
| Fundamentam. | |

#### Exploratory

### **Efficacy Endpoints**

At all efficacy assessment timepoints

- ACR 20/50/70 response rate
- Change from baseline in DAS28(ESR)
- Proportion of subjects achieving categorical DAS28(CRP) / DAS28(ESR) response (moderate/good EULAR response)
- Proportion of subjects achieving DAS28(CRP) / DAS28(ESR) remission.
- Change from baseline in Simplified Disease Activity Index (SDAI) and the Clinical Disease Activity Index (CDAI)
- Change from baseline in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue
- Note: For composite endpoints, e.g., DAS28(CRP), ACR Response, etc., each component of the
  assessment will also be reported. Results over time, reflecting all assessment time points, will also be
  reported.

#### **Biomarker Endpoints**

- Pharmacodynamic biomarkers to assess target engagement (e.g., serum concentration of free GM-CSF, GM-CSF-GSK3196165 complex)
- Pharmacodynamic biomarkers which may be predictive of response to GSK3196165 (e.g., 14-3-3η, MRP8/15, ARGS neoepitope, YKL-40)
- Pharmacodynamic biomarkers to assess response to GSK3196165 (e.g. IL-6, IL-1 $\beta$ , TNF $\alpha$ , IL-17A, IL-17F)
- Whole blood ribonucleic acid (RNA) analysis

#### Safety Biomarkers

- Biomarkers which may be indicative of lung damage (e.g. SP-D, KL-6, cholestenoic acid)
- Baseline concentrations of GM-CSF autoantibodies

### 2.3. Study Design



### 2.4. Statistical Hypotheses

The primary objective of this study is to assess the PK, safety and tolerability of GSK3196165 in combination with MTX therapy in Japanese RA subjects. No formal hypotheses to be tested. Two-sided 90% confidence interval (CI) will be used for PK estimation.

### 3. PLANNED ANALYSES

### 3.1. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. all criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG prodcedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screening | Comprise of all subjects who are given subject<br>number and of whom data are collected at<br>screening. | Study Population |
| Randomised | <ul> <li>All subjects who are randomized to treatment.</li> <li>Any subject who receives a treatment randomization number will be considered to have been randomized.</li> </ul> | Study Population |
| ITT | All subjects who are randomized to treatment and who receive at least one dose of study treatment. | Study Population |
| | | Efficacy |
| | | Safety |
| PK | This population consists of all GSK3196165-<br>treated subjects from whom PK samples are<br>collected and analyzed. | • PK |
| Immunogenicity | The immunogenicity population will consist of<br>all subjects in the ITT population, who had at<br>least one immunogenicity assessment. | Immunogenicity |

#### NOTES:

 Please refer to Appendix 10: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

• Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Time & Events |
| 11.2 | Appendix 2: Assessment Windows |
| 11.3 | Appendix 3: Treatment States and Phases |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 11.7 | Appendix 7: Multiple Comparisons & Multiplicity |
| 11.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses. |

### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Analyses

The study population analyses will be based on the All Screening, Randomised and ITT population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data | Displays Gen | erated |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition for the Subject Conclusion Record | Υ | | |
| Reasons for Subject Withdrawal | | | Υ |
| Treatment Status and Reasons for Discontinuation of Study Treatment | Υ | | Υ |
| Screening Status and Reasons for Screen Failure | Y | | Υ |
| Subjects Who Were Rescreened | | | Υ |
| Subjects Enrolled by Site ID | Υ | | |
| Subjects for Whom the Treatment Blind was Broken | | | Υ |
| Planned and Actual Treatments | | | Υ |
| Protocol Deviations | | <b>!</b> | l |
| Important Protocol Deviations | Y | | Y |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Υ |
| Populations Analysed | | | |
| Study Populations | Y | | |
| Exclusions from ITT Population | Υ | | |
| Subjects Excluded from Any Population | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y | | Υ |
| Baseline Efficacy Parameters | Υ | | |
| RF and ACPA | Υ | | Υ |
| Age Ranges | Υ | | |
| Race and Racial Combinations | Υ | | Y [1] |
| RA Disease History | Υ | | Y |
| Substance Use | Υ | | Υ |
| Prior and Concomitant Medications | | • | l |
| Medical Conditions | | | Υ |
| Medications | Υ | | Υ |
| Medications for RA prior to the Date of first dose | Υ | | |
| Medications for RA from the Date of first dose | Υ | | |
| Relationship of Medication Class, Dictionary Term and Verbatim Text | | | Y |
| Oral Corticosteroid by Visit | Υ | | |
| Change from Baseline in Oral Corticosteroid by Visit | Υ | | |
| Non-drug therapy | | | Υ |
| Exposure and Treatment Compliance | | | |
| Exposure to Study Treatment | Υ | | Υ |
| Exposure to MTX | Υ | | Υ |

### NOTES:

• Y = Yes display generated. [1] Listing of race.

### 6.1.1. Demographic Characteristics

The following items will be summarized and listed by dose group in addition to those as standard.

- BMI
- Family history for Cardiovascular risk factor

### 6.1.2. Baseline Efficacy Parameters

The following efficacy parameters at baseline will be summarized by dose group.

- DAS28(CRP, ESR)
- CRP, ESR
- Swollen Joint Count 66
- Tender Joint Count 68
- SDAI, CDAI
- Patient's Global Assessment of Arthritis
- Physician's Global Assessment of Arthritis
- Patient's Assessment of Arthritis Pain (current and past week's pain)
- HAQ-DI score
- FACIT-Fatigue

#### 6.1.3. Rheumatoid Factor and Anti-cyclic Citrullinated Protein Antibody

The number and percentage of RF positives and ACPA positives will be summarized.

#### 6.1.4. RA disease history

RA disease history will be summarized in form of disease duration categorical (< 2 years/ ≥2 years) and as summary statistics (in month), RA functional class and time since start of RA symptoms. Disease duration and time since start of RA symptoms are defined in the Appendix 5.

#### 6.1.5. Corticosteroid use

Value and change from baseline in average daily prednisolone dose will be summarized and listed by visit. Average daily dose is defined in the Appendix 5.

#### 6.1.6. Exposure

The extent of exposure to GSK3196165 and MTX will be evaluated by summarizing and listing the following items, respectively. These items are defined in the Appendix 5.

#### 6.1.6.1. GSK3196165

- The number of injections
- Cumulative dose in mg
- The duration of drug exposure in days

#### 6.1.6.2. MTX

• Overall average weekly dose

### 7. PRIMARY STATISTICAL ANALYSES

### 7.1. Pharmacokinetic Analyses

### 7.1.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the PK population, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Endpoint / Parameter/ | | Untransformed | | | | | | | Log-Transformed | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | Stats Analysis | | Sum | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Serum GSK3196165 Concentrations | | | | | | | | | | | | | | |
| Serum Concentration | | | | Υ | Υ | Υ | Υ | | | | | | | |
| PK Parameters | | | | | | | | | | | | | | |
| Parameters | | | | Υ | | | Υ | | | | Υ | | | |
| Dose Proportionality | | | | | | | | Υ | | | | Υ | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 7.1.2. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Process & Standards).

#### 7.1.3. Pharmacokinetic Parameters

### 7.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Process & Standards).
- The PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using WinNonlin (version 6.3 or higher).
- All calculations of non-compartmental parameters will be based on actual sampling times.
- PK parameters described in Table 4 will be determined from the serum GSK3196165 concentration-time data, as data permits.

Table 4 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUCtau | Area under the concentration-time curve from time zero (pre-dose in Visit 10) to 336 hr post-dose (Visit 12). |
| | If a sampling time deviation occurred at nominal time 336 hours after administration (and 336 < t), AUCtau will be calculated using the concentration at time 336 hours after administration post-dose estimated by the method of interpolation. |
| | If nominal time 336 hours after administration > t (or if the concentration at time 336 hours after administration was below then limit of quantification), then the concentration (y) at time 336 hours after administration is estimated using $\lambda z$ and last observed Ct according to the formula: y=Ct(obser) x e <sup>-<math>\lambda z(336-t)</math></sup> |
| | Then the following equation will be used to calculate (AUCtau=AUC(0-336) after last-dosing) where t is the time of last quantifiable serum concentration. AUCtau = AUC(0-t) + AUC(t-336) |
| | If $\lambda z$ is not estimable, a AUC(t-336)is not calculated (when 336 > t). (NOTE: $\lambda z$ is the apparent terminal phase rate constant.) |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose in Visit 10) to the time of the last quantifiable concentration (C(t)) will be calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). NOTE: Ct is the last observed quantifiable concentration. |
| AUC(0-inf) | Area under the concentration-time curve from time zero (pre-dose in Visit 10) extrapolated to infinity will be calculated as: AUC = AUC(0-t) + C(t) / lambda_z |
| %AUCex | The percentage of AUC(0-inf) obtained by extrapolation (%AUCex) will be calculated as: [AUC(0-inf) – AUC(0-t)] / AUC(0-inf) x 100 |

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed concentration after last dosing (Visit 10), determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| tlast | The time of the last measurable (positive) concentration. |
| t1/2 | Apparent terminal half-life will be calculated as: |
| | t1/2 = ln2 / lambda_z |
| lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the curve. |
| lambda_z_lower | The lower limit on time for values to be included in the calculation of Lambda z. |
| lambda_z_upper | The upper limit on time for values to be included in the calculation of Lambda z. |
| #pts | The number of time points used in computing Lambda z. |
| R2 | The goodness of fit statistic for the terminal elimination phase. |

#### NOTES:

Additional parameters may be included as required.

### 7.1.3.2. Statistical Analysis of Pharmacokinetic Parameters

The following PK statistical analyses will only be performed, if sufficient data is available (i.e. if subjects have well defined serum profiles).

### **Pharmacokinetic Statistical Analyses**

### **Drug Concentration Measurements**

- Summary statistics, by dose group and nominal time point, will be calculated for the concentration of GSK3196165 in serum.
- Individual serum concentration-time profiles will be plotted. Also median/mean profiles will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the loge-transformed scale (i.e. semi-log plot).
- Mean/Median profiles by dose group will be plotted. Each of figures will contain one plot on the
  untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. a loglinear plot).
- Individual subject serum concentrations of GSK3196165 will be listed by dose group and nominal time. The items to be listed are center, subject, age, sex, race, dose, date, planned relative time, actual time, time deviation, actual relative time and concentration by dose groups.

### **Deriving and Summarizing Pharmacokinetic Parameters**

- The summary tables will be produced for the derived serum GSK3196165 PK parameter. Summary statistics will be calculated for each parameter by dose groups.
- All the derived PK parameters for GSK3196165 will be listed, by subject and dose group. The
  items to be listed are center, subject, age, sex, race, dose, Cmax, Tmax, AUCtau, AUC(0-t),
  AUC(0-inf), %AUCex and t1/2.
- Individual parameter, tlast, lamda\_z, lamda\_z\_lower, lamda\_z\_upper, #pts and R2 will be listed. Summary statistics will not be calculated.
- The steady-state will be examined graphically by plotting the Ctrough of Visit 2 Visit 12 [Visit2 (Day 1), Visit4 (Day 8), Visit5 (Day 15), Visit7 (Day 29), Visit9 (Day 57), Visit10 (Day 71), Visit12 (Day 85)].

### **Pharmacokinetic Statistical Analyses**

### Dose proportionality

 Dose proportionality of GSK3196165 for Cmax, AUCtau, AUC(0-t) and AUC(0-inf) will be evaluated using the power model defined as follows.

$$log(Y_i) = \mu + \beta^* log(D_k) + \epsilon_i$$

 $Y_i$  The measured response variable of PK parameter(Cmax, AUCtau, AUC(0-t) and AUC(0-inf)) for *i*th subject

μ Intercept

β Slope of loge-transformed dose

D<sub>k</sub> Dose (k=1: 45mg, 2: 90mg, 3: 180mg)

 $\varepsilon_i$  Random error following normal distribution N(0,  $\sigma^2$ )

- The power model will be fitted to loge-transformed PK parameters data using SAS Proc Mixed with loge-transformed dose as fixed effect. An estimate of the slope with corresponding 90% CI will be estimated from the power model to assess the degree of dose-proportionality (slope β around unity indicates dose-proportionality). Point estimates for the slopes of PK parameters with associated 90% CI will be presented.
- If data permit, mean profile of Cmax, AUCtau, AUC(0-t) and AUC(0-inf) will be plotted. Each of the figures will contain one plot on linear and logarithmic scales.

### 7.2. Safety Analyses

The safety analyses will be based on the ITT population, unless otherwise specified. The summaries will be presented based on the AEs during on-treatment period. The listings will be presented based on the AEs during entire study. On-treatment is defined in the Appendix 3.

### 7.2.1. Overview of Planned Adverse Event Analyses

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 5 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | | Abso | lute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Υ | | Υ |
| All AEs by SOC and PT and Maximum Intensity | Υ | | |
| AESI | Υ | | |
| AESI – Serious Infections and Non Serious Pulmonary or Opportunistic | | | Υ |
| Infections | | | ' |
| AESI – Systemic Hypersensitivity Reactions | | | Υ |
| AESI – Injection Site Reaction | | | Υ |
| Adverse Events by Overall Frequency | Υ | | |
| Drug-Related AEs by SOC and PT | Υ | | |
| Drug-Related AEs by SOC and PT and Maximum Intensity | Υ | | |
| Common Non-Serious Adverse Events by SOC and PT | Υ | | |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Υ |
| AEs Leading to Withdrawal from Study | Υ | | |
| AEs Leading to Permanent Discontinuation of Study Treatment | Υ | | |
| AESI Leading to Permanent Discontinuation of Study Treatment | Υ | | |
| Disease Related Events | Υ | | Υ |
| Serious AEs | | | |
| Serious AEs | | | Υ |
| Serious AEs by SOC and PT | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8. SECONDARY STATISTICAL ANALYSES

### 8.1. Safety Analyses

### 8.1.1. Overview of Planned Other Safety Analyses

The safety analyses will be based on the ITT population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 6 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Ch | ange | from BL |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | | | | |
| Change from Baseline in ECG Values by Visit | | | | Υ | | |
| ECG values by Visit | Υ | | Y | | | |
| Abnormal ECG Findings | | | Υ | | | |
| Vital Signs | | | | | | |
| Change From Baseline in Vital Signs by Visit | | | | Υ | | |
| Vital Signs by Visit | Υ | | Υ | | | |
| Pulmonary | | | | | | |
| Cough by Visit and Grade | Υ | | Υ | | | |
| Lung Auscultation by Visit | Υ | | Y | | | |
| Pulse Oximetry by Visit | Υ | | Υ | Υ | | |
| Borg Dyspnea Scale by Visit | Υ | | Y | | | |
| FEV₁ by Visit | Υ | | Υ | Υ | | |
| FVC by Visit | Υ | | Y | Υ | | |
| D <sub>LCO</sub> by Visit | Υ | | Y | Υ | | |
| Respiratory events | | | | | | |
| Persistent cough with grade 2 or greater recorded | Υ | | Y | | | |
| Persistent dyspnea with grade 3 or greater recorded | Υ | | Y | | | |
| Persistent D <sub>LCO</sub> by >15% | Υ | | Y | | | |
| Hepatic B Virus | | | | | | |
| HBV DNA monitoring | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated,
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.1.1.1. Pulmonary assessment

All pulmonary assessment results (Cough, Lung Auscultation, Pulse Oximetry, Borg Dyspnea Scale, FEV<sub>1</sub>, FVC and D<sub>LCO</sub>) will be listed.

The values and the changes from baseline for the FEV<sub>1</sub>, FVC, D<sub>LCO</sub> and Pulse Oximetry will be summarized. The number and percentages of subjects having a cough for each grade and each Borg dyspnea scale will be summarized by visit.

### 8.1.1.2. Respiratory events

Numbers and percentages of subjects experiencing persistent cough, or persistent dyspnea or persistent  $D_{LCO}$  decrease will be reported in a table by dose group at the start time of the event.

The definitions of these events are described in the Appendix 5.

### 8.1.2. Overview of Planned Clinical Laboratory Analyses

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

If a subject fails any of the laboratory inclusion/exclusion criteria, laboratory test related to the inclusion/exclusion criteria may be repeated in screening period. The data collected by retests are not at screening visit but unscheduled visit. Therefore the summary at Screening visit will not be presented and baseline values defined in the Appendix 4 will be summarized.

Table 7 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Summary | | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | | | | | |
| Chemistry Changes from Baseline | | | | Υ | | |
| Chemistry by visit | Υ | | Υ | | | |
| Emergent Chemistry Results Relative to Normal Range | Υ | | | | | |
| Hematology | | | | | | |
| Hematology Changes From Baseline | | | | Υ | | |
| Hematology by Visit | Υ | | Y | | | |
| Emergent Hematology Results Relative to Normal Range | Υ | | | | | |
| Urinalysis | | | | | | |
| Urinalysis Dipstick Results | Υ | | Y | | | |
| Hepatobiliary (Liver) | | | | | | |
| Liver Monitoring/Stopping Event Reporting | | | <b>Y</b> [1] | | | |
| Hepatobiliary Laboratory Abnormalities | <b>Y</b> [1] | | | | | |
| Medical Conditions for Subjects with Liver Stopping<br>Events | | | <b>Y</b> [1] | | | |
| Substance Use for Subjects with Liver Stopping Events | | | <b>Y</b> [1] | | | |
| Liver Monitoring/Stopping Event Reporting | | | <b>Y</b> [1] | | | |
| Liver Stopping Event Information for RUCAM Score | | | <b>Y</b> [1] | | | |
| Liver Biopsy Details | | | <b>Y</b> [1] | | | |
| Liver Imaging Details | | | <b>Y</b> [1] | | | |

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Summary | | Individual |
| | Т | F | L | T | F | L |
| Laboratory Tests (Antigen and Antibody) for Liver Events | | | <b>Y</b> [1] | | | |
| Laboratory Tests (DNA and RNA) for Liver Events | | | <b>Y</b> [1] | | | |
| Cardiovascular | | | | | | |
| ECG Findings in Cardiovascular Events | | | <b>Y</b> [2] | | | |
| Subjects who had Cardiovascular Events | | | <b>Y</b> [2] | | | |
| Diagnostic Test for Cardiovascular Events | | | <b>Y</b> [2] | | | |
| Findings about Cardiovascular Events | | | <b>Y</b> [2] | | | |
| Healthcare Resource Utilization due to Cardiovascular Events | | | <b>Y</b> [2] | | | |
| NYHA Functional Class for Cardiovascular Events | | | <b>Y</b> [2] | | | |
| Death in Cardiovascular Events | | | <b>Y</b> [2] | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- RUCAM: Roussel Uclaf Causality Assessment Method
- [1]: if at least one Liver event occurs, this display will be presented.
- [2]: if at least one Cardiovascular event occurs, this display will be presented.

### 8.1.3. Immunogenicity Analyses

The immunogenicity analyses will be based on the Immunogenicity population, unless otherwise specified.

The positive subjects of Anti-GSK3196165 Binding Antibody Detection are defined as those of which tests at Confirming are "positive", and otherwise negative. The positive subjects of Neutralising Antibody detection are defined those of which tests at Screening are "positive", and otherwise negative.

The number and percentage of positive and negative subjects will be summarized. Shift table from baseline to every assessment will be produced to assess the number of subjects going from:

- negative→negative
- negative→positive
- positive→negative
- positive → positive

Anti-GSK3196165 Binding Antibody Detection (posistive/negative) will be listed together with titre value (mL) and Rheumatoid Factor (positive/negative) for each subject with at least one positive result of Anti-GSK3196165 Binding Antibody Detection.

Table 8 Overview of Immunogenicity Analyses

| [Endpoint / | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| Parameter/ Display | Stat | ts Ana | alysis | Sum | mary | Individual | |
| Type] | Т | F | L | T | F | F | L |
| Immunogenicity | | | | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.2. Efficacy Analyses

### 8.2.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the ITT population, unless otherwise specified.

Table 9 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 9 Overview of Planned Efficacy Analyses

| [Endpoint / | | Absolute | | | | | | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Stats Analysis | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | | |
| Type] | T | F | L | T | F | F | | Т | F | L | Т | F | F | L |
| DAS28 (CRP) | | | | | | | | | | | | | | |
| Values | | | | Υ | | | Υ | | | | Υ | Υ | | Υ |
| Longitudinal data analysis | | | | | | | | Υ | Υ | | | | | |
| Dose response analysis at Week 12 | | | | | | | | Υ | Υ | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.2.2. DAS28 (CRP)

DAS28(CRP) values will be listed and summarized by dose group and nominal time. Mean and Median change from baseline versus time profile by dose group will be plotted.

### 8.2.2.1. Planned Efficacy Statistical Analyses

### Statistical Analyses – Mixed Model with Repeated Measures –

### Endpoint(s)

Change from baseline in DAS28 (CRP)

### **Model Specification**

- This endpoint will be analyzed using a mixed-models repeated measures (MMRM) approach.
- Analysis will include the following fixed effects:
  - Dose group as a categorical variable
  - Visit as a categorical variable
  - Baseline DAS28(CRP) as a continuous variable
  - Dose-by-visit interaction
  - Visit-by-baseline interaction
- An unstructured variance structure will be used to model the within-patient errors.
- Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors.

### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- LSmeans for each dose will be presented along with the associated 95% CI.
- Point estimates and their associated 95% CI will be calculated for the differences between each GSK3196165 dose group and Placebo (GSK3196165 – Placebo).
- The primary treatment comparison will be the contrast between the GSK3196165 groups to placebo.

### Statistical Analyses - Dose response Analysis -

### Endpoint(s)

Change from baseline in DAS28 (CRP) at Week 12.

#### **Model Specification**

• The following non-linear models will be fitted exploratory.

$$DAS28(CRP)_{i} = E_{0} + \frac{E_{\text{max}}Dose_{i}}{Dose_{i} + ED_{50}} + \varepsilon_{i}$$

$$DAS28(CRP)_{i} = E_{0} + \frac{E_{\text{max}}Dose_{i}^{B}}{Dose_{i}^{B} + ED_{50}^{B}} + \varepsilon_{i}$$

$$DAS28(CRP)_i = E_0 + E_1 \times Dose_i + \varepsilon_i$$

- The notation in the formula is as below:
  - Subscript i denotes i-th subject.
  - E<sub>0</sub>: Response at dose 0 (placebo)
  - E<sub>max</sub>: Maximum effect (for reduction, Emax≤0; for increase, Emax≥ 0)
  - ED<sub>50</sub>: Dose at which 50% of maximum effect is reached

### Statistical Analyses - Dose response Analysis -

- B: a slope factor
- E<sub>1</sub>: Coefficient of a linear model.
- $\varepsilon_i$ : Residual error following N(0, $\sigma^2$ )
- The dose will be set to zero for all placebo data.
- Starting values for the iterations will be chosen based on the observed data as appropriate. For example;
  - E<sub>0</sub>: Mean in Placebo
  - E<sub>max</sub>: Mean difference between 180 mg and Placebo (180 mg Placebo)
  - ED<sub>50</sub>: 90 (= (180 0) / 2)
  - B = 1
- Each of the models will be fitted to the data and their fit compared using the Akaike information criteria (AIC).
- The model with the smallest AIC will be selected as the final model for inference.

### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

### Calculation procedure for the 95% CIs using a bootstrap method

- The 95% CIs will be calculated in accordance with the following procedure.
  - 1. Recreate the dataset by sampling with replacement from the original dataset by dose group.
    - Use a PROC SURVEYSELECT with SEED = 161216 to generate the bootstrap dataset
  - 2. Fit the final dose response model to the dataset in step 1. Estimate the parameters of interest  $\hat{\theta}_1$  and compute  $g(\hat{\theta}_1)$  {g is any arbitrary function.}
  - 3. Repeat steps 1-2, for b = 1, 2, ..., B (B=10,000) to obtain  $\hat{\theta}_1, \hat{\theta}_2, \ldots, \hat{\theta}_B$  and compute  $g(\hat{\theta}_1), g(\hat{\theta}_2), \ldots, g(\hat{\theta}_B)$ .
  - 4. Select 2.5% quantile of the  $\hat{\theta}_b$  and  $g(\hat{\theta}_b)$  as the lower limit and 97.5% quantile as the upper limit.

#### **Model Results Presentation**

- The result of the final model will be presented.
- The estimates of model parameters and their 95% CI will be presented.
- From the fitted model, predictive responses for each of the doses will be calculated along with 95% CI.
- The differences between each GSK3196165 dose and Placebo and their 95% CI will be calculated from the fitted model.
- A plot of the residuals versus predicted values will be examined to assess distuributional assumptions.
- The results of the other models will be shown as only SAS outputs.

### 9. EXPLORATORY STATISTICAL ANALYSES

### 9.1. Overview of Planned Exploratory Analyses

The exploratory analyses will be based on the ITT population, unless otherwise specified.

Table 10 provides an overview of the planned exploratory analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 10 Overview of Planned Exploratory Analyses

| [Endpoint / | | | Α | bsolu | te | | | | С | hange | from | Basel | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | | s Ana | lysis | Sum | mary | Indiv | idual | Sta | ts Ana | lysis | Sum | mary | Indiv | idual |
| Type] | Т | F | L | Т | F | F | L | Т | F | L | T | F | F | L |
| Efficacy Endpoints | | | | | | | | | | | | | | |
| ACR 20/50/70 response | <b>,</b> | • | 1 | 1 | | 1 | 1 | ı | 1 | 1 | 1 | 1 | 1 | |
| Proportion at each | | | | Υ | Υ | | Υ | | | | | | | |
| assessment | | | | <u> </u> | <u> </u> | | | | | | | | | |
| DAS28(ESR) | Π | I | I | | | I | | ı | Ι | I | | | I | |
| Values | | | | Υ | | | Υ | | | | Υ | Υ | | Υ |
| Longitudinal data | | | | | | | | Υ | Υ | | | | | |
| analysis | F (* | | | | | | | | | | | | | |
| SDAI, CDAI and FACIT- | Fatig | ue | I | V | 1 | I | - V | I | l | I | | | l | |
| Values | | | | Υ | | | Υ | | | | Υ | Υ | | |
| Longitudinal data | | | | | | | | Υ | Υ | | | | | |
| analysis | D) / D/ | N C 2 0 / I | CCD) . | | | | | | | | | | | |
| Categorical DAS28(CRI<br>DAS28(CRP) / DAS28(E | | | | respor | 156 | | | | | | | | | |
| Proportion at each | | | | \ \ \ | | | \ \ | | | | | | | |
| assessment | | | | Υ | | | Υ | | | | | | | |
| Other endpoints | | | | | | | | | | | | | | |
| Swollen (28, 66) & | | | | | | | | | | | | | | |
| Tender (28, 68) Joint | | | | Υ | | | Υ | | | | Υ | | | |
| Count | | | | | | | | | | | | | | |
| Patient's Assessment | | | | | | | | | | | | | | |
| of Arthritis Pain | | | | Υ | | | Υ | | | | Υ | | | |
| (current pain/past | | | | ' | | | ' | | | | ' | | | |
| week's pain) | | | | | | | | | | | | | | |
| Patient's Global | | | | Υ | | | Υ | | | | Υ | | | |
| Assessment of Arthritis | | | | <u>'</u> | | | ľ | | | | | | | |
| Physician's Global | | | | Υ | | | Υ | | | | Y | | | |
| Assessment of Arthritis | | | | I | | | I | | | | I I | | | |
| CRP, ESR | | | | Υ | | | Υ | | | | Υ | Υ | | |
| HAQ-DI score | | | | Υ | | | Υ | | | | Υ | Υ | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated, HAQ-DI: Health Assessment Questionnaire Disability Index
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 9.1.1. ACR 20/50/70 response

The number and percentage of responder will be presented. The difference of response rate from Placebo and the associated 95% CI will be calculated. The 95% CI will be based on normal approximation.

The percentage of ACR 20/50/70 responder by dose group will be plotted, respectively.

### 9.1.2. DAS28 (ESR)

DAS28(ESR) values will be listed and summarized by dose group and nominal time. Mean and median change from baseline versus time profiles by dose group will be plotted.

### Statistical Analyses – Mixed Model with Repeated Measures –

### Endpoint(s)

Change from baseline in DAS28(ESR)

#### **Model Specification**

- This endpoint will be analyzed using a MMRM approach.
- Analysis will include the following fixed effects:
  - Dose group as a categorical variable
  - Visit as a categorical variable
  - Baseline DAS28(ESR) as a continuous variable
  - Dose-by-visit interaction.
  - Visit-by-baseline interaction.
- An unstructured variance structure will be used to model the within-patient errors.
- Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Point estimates and their associated 95% CI will be calculated for the differences between each GSK3196165 dose group and Placebo (GSK3196165 Placebo).
- The primary treatment comparison will be the contrast between treatments at week 12.

### 9.1.3. SDAI, CDAI and FACIT-Fatigue

SDAI, CDAI and FACIT-Fatigue scores will be listed and summarized by dose group and nominal time. Mean and median change from baseline versus time profiles by dose group will be plotted.

### Statistical Analyses – Mixed Model with Repeated Measures –

#### Endpoint(s)

• Change from baseline in SDAI, CDAI and FACIT-Fatigue

#### **Model Specification**

This endpoint will be analyzed using a MMRM approach.

### Statistical Analyses – Mixed Model with Repeated Measures –

- Analysis will include the following fixed effects:
  - Dose group as a categorical variable
  - Visit as a categorical variable
  - Baseline as a continuous variable
  - Dose-by-visit interaction
  - Visit-by-baseline interaction
- An unstructured variance structure will be used to model the within-patient errors.
- Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors.

### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- LSmeans for each dose will be presented along with the associated 95% CI.
- Point estimates and their associated 95% CI will be calculated for the differences between each GSK3196165 dose group and Placebo (GSK3196165 – Placebo).

### 9.1.4. Categorical DAS28 Response

A good or moderate response will be combined to form the "responder" category. The number and percentage of responders will be presented. The difference of response rate from Placebo and the associated 95% CI will be calculated. The 95% CI will be based on normal approximation.

#### 9.1.5. DAS28 Remission

The number and percentage of remission from Placebo will be presented. The difference of remission rate and the associated 95% CI will be calculated. The 95% CI will be based on normal approximation.

#### 9.1.6. Other endpoints

The other endpoints as below will be listed and summarized by dose group and nominal time as well as changes from baseline. Changes from baseline in only CRP, ESR and HAQ-DI will be plotted by dose group, respectively.

- Swollen Joint Count (28 and 66)
- Tender Joint Count (28 and 68)
- Patient's Assessment of Arthritis Pain
  - Current pain
  - Past week's pain
- Patient's Global Assessment of Disease Activity
- Physician's Global Assessment of Arthritis

- CRP (in mg/L), ESR (in mm/hr)
- Health Assessment Questionnaire-Disability Index (HAQ-DI)

### 9.2. Pharmacodynamic and Biomarker Analyses

### 9.2.1. Overview of Planned Pharmacodynamic and Biomarker Analyses

The pharmacodynamic analyses will be based on the ITT population, unless otherwise specified.

Table 11 provides an overview of the planned pharmacodynamic and Biomarker analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 11 Overview of Planned Pharmacodynamic and Biomarker Analyses

| Endpoint / Parameter/ | Untransformed | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Display Type | | | A | bsolu | ite | | Change from Baseline | | | | | | | |
| | Stat | s Ana | lysis | Sum | mary | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Т | F | L | T | F | F | L | Т | F | L | T | F | F | L |
| free soluble GM-CSF and soluble GM-CSF complexed to GSK3196165 | | | | | | | | | | | | | | |
| Values | | | | Υ | Υ | | Υ | | | | Υ | Υ | | Υ |
| MRP8/14, ARGS neoepi | tope, | YKL- | 40 an | d 14-3 | -3η. | | | | | | | | | |
| Values | | | | Υ | Υ | | Υ | | | | Υ | Υ | | Υ |
| IL-6, IL-1β, TNFα, IL-17/ | A and | IL-17 | F | | | | | | | | | | | |
| Values | | | | Υ | Υ | | Υ | | | | Υ | Υ | | Υ |
| SP-D, KL-6 and cholest | enoic | acid | | | | | | | | | | | | |
| Values | | | | Υ | Υ | | Υ | | | | Υ | Υ | | Υ |
| measurement of GM-CS | SF au | toanti | bodie | s at b | aselin | е | | | | | | | | |
| Values | | | | Υ | | | Υ | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

Biomarkers/pharmacodynamic endpoint values will be listed and summarized by dose group and nominal time. Mean and median versus time profiles by dose group will be plotted.

### 9.3. Pharmacokinetic / Pharmacodynamic Analyses

A graphical PK/PD exploration will be conducted to complement the statistical doseresponse analysis and to visualize the nature of the concentration-response correlation. A variety of graphs will be generated per subject and in overall, where GSK3196165 concentration is characterised by the individual values, and the response is characterised by the individual values of the pharmacodynamic markers or efficacy.

#### CONFIDENTIAL

201789

Pharmacokinetic and pharmacodynamic data from this study may be combined with historical data (e.g. BAROQUE) for the purpose of further exploratory analysis (including population pharmacokinetic and/or PK/PD modelling as appropriate) which may be reported separately from the main clinical study report.

- Linear scatterplot of change from baseline in PD values (free soluble GM-CSF, GM-CSF-GSK3196165 complex) at each visit versus GSK3196165 concentration values at corresponding visit
- Linear scatterplot of change from baseline in CRP levels at each visit versus GSK3196165 concentration values at corresponding visit
- Linear scatterplot of change from baseline in DAS28(CRP) measures at each visit versus GSK3196165 concentration values at corresponding visit

### 10. REFERENCES

Aletaha D, Nell VP, Stamm T, et al. Acute phase reactants add little to composite disease activity indices for rheumatoid arthritis: validation of a clinical activity score. *Arthritis Res Ther.* 2005;7(4):R796-806.

American Collenge of Rheumatology Committee to Reevaluate Improvement Criteria. A proposed revision to the ACR20: the hybrid measure of American College of Rheumatology response. *Arthritis Rheum.* 2007;57(2):193-202.

Fransen J, van Riel PL,. The Disease Activity Score and the EULAR response criteria. *Clin Exp Rheumatol.* 2005;23(5 Suppl 39):S93-9.

Fries JF, Spitz P, Kraines RG, et al. Measurement of patient outcome in arthritis. *Arthritis Rheum.* 1980;23(2):137-45.

GlaxoSmithKline Document Number 2016N278580\_01: Study Protocol of 201789: A Phase 1/2, Double-Blind, Placebo-Controlled Study of the Pharmacokinetics, Safety and Tolerability of GSK3196165 in Combination with Methotrexate Therapy, in Japanese Subjects with Active Moderate-Severe Rheumatoid Arthritis Despite Treatment with Methotrexate. Effective Date- 26-Sep-2016.

Matsuda Y, Singh G, Yamanaka H, et al. Validation of a Japanese Version of the Stanford Health Assessment Questionnaire in 3,763 Patients With Rheumatoid Arthritis. *Arthritis & Rheumatism.* 2003;49(6):784-8.

Prevoo ML, van't Hof MA, Kuper HH, et al. Modified disease activity scores that include twenty-eight joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. *Arthritis Rheum.* 1995;38(1):44-8.

Smolen JS, Breedveld FC, Schiff MH, et al. A simplified disease activity index for rheumatoid arthritis for use in clinical practice. *Rheumatology (Oxford)*. 2003;42(2):244-57.

Wells G, Becker JC, Teng J, et al. Validation of the 28-joint Disease Activity Score (DAS28) and European League Against Rheumatism response criteria based on C-reactive protein against disease progression in patients with rheumatoid arthritis, and comparison with the DAS28 based on erythrocyte sedimentation rate. *Ann Rheum Dis.* 2009;68(6):954-60.

### 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 11.1 | Appendix 1: Time and Events |
| Section 11.2 | Appendix 2: Assessment Windows |
| Section 11.3 | Appendix 3: Treatment States & Phases |
| Section 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | <ul> <li>Study Treatment &amp; Sub-group Display Descriptors</li> </ul> |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.5 | Appendix 5: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Immunogenicity |
| Section 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 11.7 | Appendix 7: Multiple Comparisons and Multiplicity |
| Section 11.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 11.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 11.10 | Appendix 10: List of Data Displays |

# 11.1. Appendix 1: Time & Events

### 11.1.1. Protocol Defined Time & Events

| | Screen-<br>ing | Base | eline | | | | | | | | | | | U | Last Visit | EW <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | | | | | | | | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | |
| Procedures | Week | | | | | | | | | | | | | | | |
| | (up to 4 weeks) | 0 | | 1 | 2 | 3 | 4 | 6 | 8 | 1 | 0 | 12 | 15 | 18 | 22 | |
| | | | | | | | | D | ay | | | | | | | |
| | | 1 | 3* | 8 | 15 | 22 | 29 | 43 | 57 | 71 | 74* | 85 | 106 | 127 | 155 | |
| Allowance | | | | | ±1 day | | | ±3 days | | | ±1 day | ±3 days | ±1 week | | | |
| Written Informed Consent(s) | Χ | | | | | | | | | | | | | | | |
| Subject Demography | Χ | | | | | | | | | | | | | | | |
| Medical, Disease, Therapy History | Χ | | | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | Χ | | | | | | | | | | | | | | | |
| Efficacy and PRO Assessments <sup>3</sup> | | | | | | | | | | | | | | | | |
| Swollen (66) & Tender (68) Joint Count <sup>2</sup> | Χ | X <sup>4</sup> | | Х | Х | | Х | Х | Х | | | Х | | | Х | Х |
| Patient's Assessment of Arthritis Pain,<br>Patient's Global Assessment of<br>Arthritis, Physician's Global<br>Assessment of Arthritis <sup>3</sup> | Х | X <sup>4</sup> | | Х | Х | | Х | Х | Х | | | Х | | | Х | Х |
| HAQ-DI <sup>3</sup> | Χ | X <sup>4</sup> | | Х | Х | | Х | Х | Х | | | Х | | | Х | Χ |
| FACIT-Fatigue <sup>3</sup> | | X <sup>4</sup> | | | | | Χ | | | | | Х | | | Χ | Χ |

| | Screen-ing | Base | eline | | | | Tre | atment Pe | riod | | | | FU | | Last Visit | EW <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | | | | | | | | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | |
| Procedures | Week | | | | | | | | | | | | | | | |
| | (up to 4 weeks) | ( | ) | 1 | 2 | 3 | 4 | 6 | 8 | 1 | 0 | 12 | 15 | 18 | 22 | |
| | Day | | | | | | | | | | | | | | | |
| | | 1 | 3* | 8 | 15 | 22 | 29 | 43 | 57 | 71 | 74* | 85 | 106 | 127 | 155 | |
| Allowance | | | | | ±1 day | | | | ±3 days | | ±1 day | ±3 days | ±1 week | | | |
| Safety Evaluations <sup>5</sup> | | | | | | | | | | | | | | | | |
| Concomitant Medication | Χ | Χ | | T | T | • | | Record | all concor | mitant med | ications | | | T | | |
| Height <sup>6</sup> , Body weight | Χ | | | | | | Χ | | | | | Χ | | | Х | Х |
| Other Physical Examination <sup>7</sup> | Χ | X <sup>4</sup> | | Х | Х | | Χ | | Х | | | Χ | | | Х | Х |
| Vital Signs | Х | Х | | Х | Х | Х | Х | Х | Х | Х | | Х | | | Х | Х |
| 12-lead ECG8 | Х | | | | | | | | | | | Х | | | | Х |
| AEs/SAEs/AESIs | <b>X</b> 9 | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х | Χ | Χ |
| Cough, Lung Auscultation, Pulse Oximetry, | Х | X <sup>4</sup> | | X | х | Х | X | Х | X | X | | Х | | | Х | Х |
| Borg Dyspnea Scale | ^ | Λ | | ^ | ^ | ^ | ^ | ^ | ^ | ^ | | ^ | | | ^ | ^ |
| Chest X-ray <sup>10</sup> | Χ | | | | | | | | | | | | | | | |
| Spirometry (FEV <sub>1</sub> , FVC) | Χ | | | | | | | | | | | Χ | | | Χ | Χ |
| D <sub>LCO</sub> | X <sup>11</sup> | | | | | | | | | | | Χ | | | Χ | Χ |
| Laboratory Assessments | | | | | | | | | | | | | | | | |
| Hematology, Chemistry (except for lipid and pregnancy test) | Х | X <sup>4</sup> | | | Х | | Х | | Х | | | Х | | | Х | Х |

| | Screen-ing | Base | eline | Treatment Period | | | | | | | | | | U | Last Visit | EW <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | | | | | | | | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | |
| Procedures | Week | | | | | | | | | | | | | | | |
| | (up to 4<br>weeks) | ( | ) | 1 | 2 | 3 | 4 | 6 | 8 | 1 | 10 12 | | 15 | 18 | 22 | |
| | Day | | | | | | | | | | | | | | | |
| | | 1 | 3* | 8 | 15 | 22 | 29 | 43 | 57 | 71 | 74* | 85 | 106 | 127 | 155 | |
| Allowance | | | | 1 | ±1 day | 1 | ı | | ±3 days | ı | ±1 day | ±3 days | | ±1 week | | |
| Urinalysis (dip stick) | Χ | | | | | | Χ | | Х | | | Χ | | | Χ | Χ |
| Cholesterol, triglycerides, HDL, LDL <sup>12</sup> | | X <sup>4</sup> | | | | | | | | | | Х | | | Х | Х |
| Pregnancy test <sup>13</sup> | S | U | | | | | U | | U | | | U | | | U | U |
| TB, HBsAg, HepB cAb, HBs Ab, HepC<br>Ab, HIV, HBV DNA** | Χ | | | | | | | | | | | | | | | |
| HBV DNA monitoring (HBs Ab positive subject only) | | | | | | | X | | Х | | | Х | Х | Х | Χ | Х |
| RF, ACPA (anti-CCP) | Χ | | | | | | | | | | | | | | | |
| ESR <sup>14</sup> | | X <sup>4</sup> | | Х | Х | | Χ | Χ | Х | | | Χ | | | Χ | Х |
| CRP | Χ | X <sup>4</sup> | | Х | Χ | | Χ | Χ | Χ | | | Χ | | | Χ | Х |
| Other Laboratory Assessments | | | | | | | ı | | | r | | | | | | |
| PK blood sampling (GSK3196165) <sup>15</sup> | | X <sup>4</sup> | Х | Х | Х | | Х | | Х | Х | Х | Х | Χ | Х | Х | Χ |
| Free GM-CSF, GM-CSF-GSK3196165 complex | | X <sup>4</sup> | Х | Х | Х | | Х | | Х | Х | | Х | | | Х | Х |
| PD blood biomarkers | | X <sup>4</sup> | | | Х | | Х | | | | | Х | | | | Χ |
| RNA blood biomarker | | X <sup>4</sup> | | | | | | | | | | Х | | | Х | Х |

| | Screen-ing | -<br>Baseline | | | Treatment Period | | | | | | | | | FU | | EW <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | | | | | | | | | | |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | |
| Procedures | Week | | | | | | | | | | | | | | | |
| | (up to 4 weeks) | 0 | | 1 | 2 | 3 | 4 | 6 | 8 | 10 | | 12 | 15 | 18 | 22 | |
| | | Day | | | | | | | | | | | | | | |
| | | 1 | 3* | 8 | 15 | 22 | 29 | 43 | 57 | 71 | 74* | 85 | 106 | 127 | 155 | |
| Allowance | | | | | ±1 day | | | ±3 days ±1 | | | | ±3 days | ±1 week | | | |
| PGx sampling DNA <sup>16</sup> | | X <sup>4</sup> | | | | | | | | | | | | | | |
| Lung biomarkers | | X <sup>4</sup> | | | | | | | | | | Χ | | | Х | Χ |
| Immunogenicity (anti-GSK3196165<br>antibody) <sup>17</sup> | | X <sup>4</sup> | | | Х | | Х | | | | | Х | | | Х | Х |
| Anti-GM-CSF auto-antibodies | | X <sup>4</sup> | | | | | | | | | | | | | | |
| Study Treatment<br>GSK3196165/placebo <sup>18</sup> | | Χ | | Х | Х | Х | Х | Х | Х | Х | | | | | | |

ACPA: Anti-cyclic citrullinated protein antibody, CCP: Cyclic citrullinated peptide, ESR: Erythrocyte sedimentation rate, FVC: Forced vital capacity, HBV: Hepatitis B virus, HDL: High-density lipoprotein, LDL: Low-density lipoprotein, RF: Rheumatoid factor.

(12 weeks after last dose of study medication).

- 2. The same individual (where possible) should perform all disease assessments for an individual subject.
- 3. PRO assessments should be conducted before any tests, procedures, assessments or consultations, to avoid influencing the subjects' perception.
- 4. Assessments may be performed up to 24hours before dosing GSK3196165/placebo.
- 5. All safety evaluations should be conducted before dosing GSK3196165/placebo.
- 6. Height will be measured at only screening.
- 7. Complete physical at screening, and then limited physical examination (see Section 7.4.7 in the Protocol) thereafter.

<sup>1.</sup> All subjects who withdraw from the study should have an early withdrawal (EW) visit as soon as possible after study agent discontinuation and then return for a follow-up visit (the last visit) for 10 weeks

- 8. ECG should be performed before vital signs, blood draws, and dosing (triplicate ECGs required at screening, and single thereafter unless there are safety concerns, in which case repeats may be required
  - (see Section 7.4.9 in the Protocol).
- 9. Only SAEs related to study participation or related to a GSK product will be recorded from the time a subject consents to participate in the study.
- 10. Unless performed within previous 12 weeks (No need to repeat if subject re-screened).
- 11. Chest HRCT if D<sub>LCO</sub> ≥60% <70% predicted (No need to repeat if subject re-screened).
- 12. ≥8 hours fasting required before blood draw.
- 13. For women of child-bearing potential. S=serum; U=urine.
- 14. ESR measured locally.
- 15. PK sampling should be collected before dosing at the visits scheduled study treatment (GSK3196165/placebo). At the visits doesn't scheduled study treatments, it may be collected in any time during the
  - visit. (Day 3, 74, 85, 106, 127, 155, and early withdrawal visit).
- In consenting subjects.
- 17. In addition to these scheduled immunogenicity assessments, "event-driven" testing will also be employed for those subjects that experience anaphylaxis, serious hypersensitivity, or AEs related
  - to study drug administration that led to withdrawal from the study (see Section 7.5 in the Protocol).
- 18. GSK3196165 or placebo must be administered on the same day each week ±1 day for the first 5 weekly doses, thereafter on the same day EOW ±3 days for bi-weekly doses.
- \* The Day 3 (Visit 3) blood sample must be drawn 2 days (±1 day is allowable) after the first dose, and the Day 74 (Visit 11) blood sample must be drawn 3 days (±1 day is allowable) after the last dose.
- \*\* HBV-DNA sample will be collected from all subjects, and HBV-DNA will be tested for only subjects with HBs Ab positive.
# 11.2. Appendix 2: Assessment Windows

Data at the scheduled visit defined by Appendix 1 will be summarized according to this RAP. Data out of the allowances will not be slotted to a particular time point, but will be listed as unscheduled and early withdrawal unless otherwise specified.

In case that the one allowance contains more than two assessments, the first assessment will be treated as the scheduled and the others as the unscheduled.

### 11.3. Appendix 3: Treatment States and Phases

# 11.3.1.1. Treatment States for Concomitant Medications for Rheumatoid Arthritis (CONMEDS RA) Data



## 11.3.1.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-treatment | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 12 weeks |
| Post-treatment | AE Start Date > Study Treatment Stop Date + 12 weeks |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date, = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date, = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| Onset Time<br>Since last Dose<br>(Days) | If Treatment Stop Date > AE Onset Date, = AE Onset Date - Treatment Stop Date If Treatment Stop Date ≤ AE Onset Date, = AE Onset Date - Treatment Stop Date + 1 Missing otherwise |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship to GSK3196165/Placebo is marked 'YES' on Inform/CRF OR value is missing. |
| MTX-related | If relationship to Methotrexate is marked 'YES' on Inform/CRF OR value is missing. |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 11.4. Appendix 4: Data Display Standards & Handling Conventions

#### 11.4.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order [1] |
| Α | Placebo | Placebo | 1 |
| В | GSK3196165 45 mg | GSK3196165 45 mg | 2 |
| С | GSK3196165 90 mg | GSK3196165 90 mg | 3 |
| D | GSK3196165 180 mg | GSK3196165 180 mg | 4 |

#### NOTES:

#### 11.4.2. Baseline Definition & Derivations

#### 11.4.2.1. Baseline Definitions

For all endpoints (expect as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

#### 11.4.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 11.4.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 11.4.3. Reporting Process & Standards

| Reporting Process | |
|-------------------|------------------------------------------------|
| Software | |
| The currently sup | ported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : arenv\arprod\gsk3196165\mid201789\final_02 |
| QC Spreadsheet | :arenv\arprod\gsk3196165\mid201789\final_02\qc |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

#### **Reporting Process**

#### **Analysis Datasets**

- Analysis datasets will be created according to Legacy GSK A&R dataset standards OR CDISC standards (SDTM IG Version 3.1.3 & AdaM IG Version 1.0.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will not be generated.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the randomized group the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables, except for the Respiratory events and the laboratory items which may be re-tested.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Reporting Standards | |
|---|---|
| <b>Descriptive Summa</b> | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharm | acokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and [between and or within] geometric coefficient of variation (CVb/w (%)) will be reported.</li> <li>[1] CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data)</li> </ul> |
| Parameters Not | Tmax |
| Being Log | |
| Transformed | |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from randomization date :
  - Ref Date = Missing
     → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### 11.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be calculated based on date of Screening visit as an Age reference date for Screen failed subjects and based on date of the initial dose date for ITT population.

#### Age Group

- The following category will be used for Summary of Demography.
  - Age  $\leq$  18 (years)
  - o 19 < Age < 64
  - $\circ$  65  $\leq$  Age

#### Age Category

- The following category will be used for Summary of Age Ranges.
  - Age < 18 (years)</li>
  - $\circ$  18  $\leq$  Age  $\leq$  64
  - $\circ$  65  $\leq$  Age  $\leq$  84
  - $\circ$  85  $\leq$  Age

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Demographics**

#### RA disease history

#### **RA Disease Duration**

RA disease duration will be calculated based on the formula:

Disease Duration in Months = [Treatment Start Date – (RA Diagnosis Date)] / 30.25 rounded to four decimals

Disease Duration in Years = [Treatment Start Date – (RA Diagnosis Date)] / 365.25 rounded to four decimals

#### Time since start of RA symptoms

• Time since start of RA symptoms will be calculated based on the formula:

Time since start of RA symptoms in Months = [Treatment Start Date – (Date of first symptom)] / 30.25 rounded to four decimals

#### **Prior and Concomitant Medications**

#### **Oral Corticosteroid**

- To assess corticosteroid use and determine average daily corticosteroid dose, all corticosteroid dosages will be converted to a prednisolone equivalent in milligrams by multiplying the dose of the steroid (using the coded term from GSKDrug) by the conversion factor to get prednisolone equivalent units.
- The following table will provide the conversion factors.
- For each scheduled visit, the average daily prednisolone dose will be calculated by summing all
  prednisolone doses since the previous visit up to and including the current visit and then
  dividing by the number of days in this period (Date of current visit Date of previous
  scheduled visit).
- If frequency that a subject takes the steroid is less than once daily such as QOD, the dosage will be converted to daily dose and then the average daily dose will be calculated. For example, if a subject takes 10 mg of the steroid QOD, the daily dose is 5 mg/day.

| Conversion | Steroid |
|------------|--------------------|
| 8.333 | BETAMETHASONE |
| 0.2 | CORTISONE |
| 6.667 | DEXAMETHASONE |
| 0.25 | HYDROCORTISONE |
| 1.25 | METHYLPREDNISOLONE |
| 1 | PREDNISOLONE |
| 1.25 | TRIAMCINOLONE |

#### Rheumatoid factor (RF)

- A subject who has a value of RF > 15 IU/mL is positive.
- Otherwise negative.

### Anti-cyclic Citrullinated Protein Antibody (ACPA)

- A subject who has a value of ACPA ≥ 4.5 U/mL is positive.
- Otherwise negative.

#### **Extent of Exposure**

#### GSK3196165

• Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### Cumulative Dose = Sum of (Actual Volume x One Dosage / Expected Volume)

The following table provides the one dosage and the expected volume in each dose group.

| Dose group | One Dosage (mg) | Expected volume (mL) |
|------------|-----------------|----------------------|
| Placebo | 0 | 0.6 |
| 45 mg | 45 | 0.3 |
| 90 mg | 90 | 0.6 |
| 180 mg | 180 | 1.2 |

#### Methotrexate (MTX)

 Overall Average Weekly MTX dose will be averaged across Week 1 - 12for each subject based on the formula:

Overall Average Weekly MTX Dose = Mean of the Weekly Dosage of MTX

#### 11.5.3. Safety

Adverse events of special interest will be derived using Common Terminology Criteria for Adverse Events, 2009 v4.0 (CTCAE).

#### **Adverse Events of Special Interest**

Adverse Events of Special Interest are defined as the AEs below. AESI will be specified by Safety Review Team and Japan EST.

- Serious infections, including serious respiratory infections and TB.
- Opportunistic infections
- Neutropenia
- Respiratory events as AESI
- Pulmonary alveolar proteinosis
- Hypersensitivity reactions, including anaphylaxis
- Injection site reactions

| Respiratory events | |
|---|---|
| Events | Definition |
| Persistent cough with Grade 2 or greater recorded | Cough grade 2 or greater recorded for 3 consecutive weeks (15 or more days) on the eCRF page. |
| Persistent dyspnea with Grade 3 or greater recorded | Borg Scale grade 3 or greater recorded for 3 consecutive weeks (15 or more days) on the eCRF page. |

| Respiratory events | |
|---|---|
| Events | Definition |
| Persistent decrease of D <sub>LCO</sub> by > 15% | Relative decrease of D <sub>LCO</sub> of >15% compared to baseline for 3 consectuvie weeks (15 or more days) Decrease of D <sub>LCO</sub> = (%change from baseline in D <sub>LCO</sub> ) ×-1 A subject's baseline D <sub>LCO</sub> value will be taken as the lowest value obtained from the Screening assessment or any unscheduled visit in between Screening and Day 1 visit. |
| Final adjudication will be conducted by the SRT. | |

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
- Example 1: 2 Significant Digits = '< x ' becomes x 0.01
- Example 2: 1 Significant Digit = '> x' becomes x + 0.1
- Example 3: 0 Significant Digits = '< x' becomes x 1</p>

#### 11.5.4. **Efficacy**

**ACR 20/50/70 response**[American Collenge of Rheumatology Committee to Reevaluate Improvement Criteria, 2007]

#### **Procedure**

- The following 7 ACR-core set measures will define ACR20/50/70 response.
  - Tender/Painful Joint Count 68 (TJC68)
  - Swollen Joint Count 66 (SJC66)
  - Patient's Assessment of Arthritis Pain at this time
  - Patient's Global Assessment of Arthritis
  - Physician's Global Assessment of Arthritis
  - C-reactive protein (CRP) (in mg/L)
  - Health Assessment Questionnaire-Disability Index (HAQ-DI)
- The %Change from Baseline in each ACR-core set measure will be calculated.
- If %Change from Baseline in both tender and swollen joint counts are less than -20% and those in 3 of the 5 remaining ACR-core set measures are less than -20%, ARC20 criteria is met.
- Similarly ACR50 and 70 are calculated with the respective percent improvement.
- For all visits if any of the component scores are missing, then those scores will considered as not having met the criteria for improvement. Therefore, if TJC68 or SJC66 or 3 or more of the 5 remaining ACR-core set measures are missing, ACR20/ ACR50/ ACR70 will each be considered as "no response"
- For component scores with missing Baseline values or a Baseline value of 0, the percentage improvement cannot be calculated and the component will be considered as not having met the criteria for improvement for all visits.

# **Flowchart** Calculate %change from baseline of a subject in 7 specific components of the ACR assessments 7 components 1. Tender/Painful Joint Count (68) 2. Swollen Joint Count (66) 3. Patient's Assessment of Arthritis Pain 4. Patient's Global Assessment of Arthritis 5. Physician's Global Assessment of Arthritis 6. CRP 7. Health Assessment Questionnaire-Disability Index (HAQ-DI) . %changes from baseline in tender and swollen joint count $\leq -X$ ➤ The subject did not meet the criteria for ACRX Yes %changes from baseline in 3 of the 5 remaining components $\leftarrow$ X The subject did not meet the criteria for ACRX Yes No The subject met the criteria for ACRX

#### **Examples**

The subject did not met the criteria for ACR20

| Component | Baseline | Post-dose visit value | %change |
|---|---|---|---|
| TJC68 | 43 | 14 | -67 |
| SJC66 | 38 | 44 | 16 |
| Patient's Assessment of Arthritis Pain | 46 | 20 | -57 |
| Patient's Global<br>Assessment of Arthritis | 85 | 31 | -64 |
| Physician's Global<br>Assessment of Arthritis | 75 | 27 | -64 |
| CRP | 2.8 | 2.0 | -29 |
| HAQ-DI | 11.6 | 7.2 | -38 |

• The subject met the criteria for ACR50 but not ACR70

| Component | Baseline | Post-dose visit value | %change |
|---|---|---|---|
| TJC68 | 43 | 14 | -67 |
| SJC66 | 38 | 14 | -63 |
| Patient's Assessment of Arthritis Pain | 46 | 10 | -78 |
| Patient's Global<br>Assessment of Arthritis | 85 | 31 | -64 |
| Physician's Global<br>Assessment of Arthritis | 75 | 27 | -64 |
| CRP | 2.8 | 1.0 | -64 |
| HAQ-DI | 11.6 | 1.2 | -90 |

#### Disease Activity Score[Prevoo, 1995; Fransen, 2005; Wells, 2009]

- The DAS assessment is a derived measurement with differential weighting given to each component. The DAS28 (CRP) and DAS28 (ESR) will be calculated at each assessment time point.
- The components of the DAS28 arthritis assessment include:
  - Tender Joint Count 28 (TJC28)
  - Swollen Joint Count 28 (SJC28)
  - C-reactive protein (CRP) (in mg/L) or Erythrocyte sedimentation rate (ESR) (in mm/hr)
  - Patient's Global Assessment of Arthritis (PtGA) (visual analogue scale with values from 0 = best to 100 = worst)

#### DAS28 (CRP)

• The DAS28 (CRP) will be calculated using the following formula:

$$DAS28(CRP) = 0.56 \times \sqrt{TJC28} + 0.28 \times \sqrt{SJC28} + 0.36 \times \ln(CRP + 1) + 0.014 \times PtGA + 0.96$$

 If one of the components is missing at an individual assessment point, the DAS28 (CRP) value for that assessment will be set to missing

#### DAS28 (ESR)

The DAS28 (ESR) will be calculated using the following formula:

$$DAS28(ESR) = 0.56 \times \sqrt{TJC28} + 0.28 \times \sqrt{SJC28} + 0.70 \times \ln(ESR) + 0.014 \times PtGA$$

 If one of the components is missing at an individual assessment point, the DAS28 (ESR) value for that assessment will be set to missing. An ESR value of 0 will be substituted with ESR = 1 for the calculation of DAS28 (ESR).

#### **Categorical DAS28 Response**

- DAS28 (CRP) and DAS28 (ESR) will be categorized using EULAR response criteria.
   Response at a given time point is defined based on the combination of current DAS28 score and DAS28 decrease from baseline. The definition of no response, moderate response and good response is captured in the following table:
- DAS28 decrease from baseline value will be calculated using the following formula:

#### DAS28 decrease from baseline = DAS28 Baseline - Post-Dose Visit DAS28 Value

| Current DAC20 | DAS28 decrease from baseline | | |
|---|---|---|---|
| Current DAS28 | >1.2 | >0.6 to ≤1.2 | ≤0.6 |
| ≤3.2 | Good response | Moderate response | No response |
| >3.2 to ≤5.1 | Moderate response | Moderate response | No response |
| >5.1 | Moderate response | No response | No response |

 If the post-baseline DAS28 (CRP) or DAS28 (ESR) is missing, then the corresponding EULAR category will be missing.

#### **DAS28 Remission**

- DAS28 (CRP) remission is achieved by a DAS28 (CRP) value lower than 2.6.
- DAS28 (ESR) remission is achieved by a DAS28 (ESR) value lower than 2.6.
- Missing DAS28 values will be considered as not achieving remission.

#### Health Assessment Questionnaire-Disability Index (HAQ-DI)[Fries, 1980; Matsuda, 2003]

#### **Procedure**

- The functional status of the subject will be assessed by means of the Disability Index of the Health Assessment Questionnaire. This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in eight functional areas:
  - Dressing & grooming
  - Arising
  - Eating
  - Walking
  - Hygiene

- Reach
- Grip
- Activities
- Each functional area contains at least two questions. For each question, there is a four level response set that is scored from 0 (without any difficulty) to 3 (unable to do). If aids or devices or physical assistance are used for a specific functional area and the maximum response of this functional area is 0 or 1, the according value is increased to a score of 2.

| Aid or device | Functional area |
|-------------------------------------|-----------------------|
| Devices used for dressing | Dressing and grooming |
| Special or built up chair | Arising |
| Built up or special utensils | Eating |
| Cane | Walking |
| Crutches | Walking |
| Walker | Walking |
| Wheelchair | Walking |
| Bathtub seat | Hygiene |
| Bathtub bar | Hygiene |
| Raised toilet seat | Hygiene |
| Long-handled appliances in bathroom | Hygiene |
| Long-handled appliances for reach | Reach |
| Jar opener | Grip |

- Regarding these corrections, the highest response within each functional area determines the score of that specific functional area. If no questions within a given functional area were answered, no score will be provided for that category (even if answers on aids or equipment are available).
- HAQ-DI is only calculated if there are at least 6 functional area scores available.
- The average of these non-missing functional area scores defines the continuous HAQ-DI score ranging from 0 to 3. If there are less than 6 functional area scores available, no imputation will be done and the HAQ-DI will be set to missing for the according assessment.



### **Examples**

| estion |
|--------|

| No. | Functional area | Value |
|-----|-----------------------|-------|
| 1 | Dressing and grooming | 1 |
| 2 | Dressing and grooming | 0 |
| 3 | Arising | 2 |
| 4 | Arising | 1 |
| 5 | Eating | 3 |
| 6 | Eating | 0 |
| 7 | Eating | 2 |
| 8 | Walking | 1 |
| 9 | Walking | 0 |
| 10 | Hygiene | 2 |
| 11 | Hygiene | 2 |
| 12 | Hygiene | 1 |
| 13 | Reach | 0 |
| 14 | Reach | 0 |
| 15 | Grip | 3 |
| 16 | Grip | 2 |
| 17 | Grip | 0 |
| 18 | Activities | 2 |
| 19 | Activities | 1 |
| 20 | Activities | 0 |

### Use of aid or device / Need for help

| Functional area | Use or Need |
|-----------------|-------------|
| Dressing and | × |
| grooming | ^ |
| Arising | 0 |
| Eating | × |
| Walking | 0 |
| Hygiene | × |
| Reach | 0 |
| Grip | × |
| Activities | × |



# Maximum value in each functional area

| Functional area | Score | Use of aid | Updated score |
|---|---|---|---|
| Dressing and grooming | 1 | х | 1 |
| Arising | 2 | 0 | 2 |
| Eating | 3 | × | 3 |
| Walking | 1 | 0 | 2 |
| Hygiene | 2 | × | 2 |
| Reach 0 | | 0 | 2 |
| Grip | Grip 3 × | | |
| Activities | Activities 2 × | | |
| | Sum updated scores 17 | | |
| Divide by number of functional area scored 2.125 | | | |

This score was not updated because it was more than 2

This score was increased to 2 because it was 0 or 1.

#### **FACIT-Fatigue**

#### **Procedure**

- The FACIT-Fatigue questionnaire is a patient-reported measure developed to assess fatigue consisting 13 statements regarding feeling fatigue using a numeric rating scale ranging from 0 (Not at all) to 4 (very much).
- For only two of the items (i.e. An5 and An7) a higher value represents a lower fatigue, 11 of the item scores (i.e. HI7, HI12, An1, An2, An3, An4, An8, An12, An14, An15, An16) have to be reversed by subtracting the captured value from 4 (0 is turned to a 4, 1 into 3, 3 into 1, 4 into 0).
- After performing the reversals, the sum of the non-missing individual items will be multiplied by 13 and divided by the number of the non-missing individual items.
- The final score ranges from 0 to 52 with higher values representing a lower fatigue.
- If more than 6 individual items are missing at an assessment the FACIT-Fatigue score will be set to missing at that assessment.

#### **Examples**

| Item Code | Reverse Ite | m | Item Respons | е | Item Score |
|-----------|-------------|----------|--------------------|------|------------|
| HI7 | 4 | <u> </u> | 2 | = | 2 |
| HI12 | 4 | <u> </u> | 4 | = | 0 |
| An1 | 4 | <u> </u> | 3 | = | 1 |
| An2 | 4 | - | 1 | = | 3 |
| An3 | 4 | <u> </u> | 3 | = | 1 |
| An4 | 4 | <u> </u> | 0 | = | 4 |
| An5 | 0 | + | 2 | = | 2 |
| An7 | 0 | + | 1 | = | 1 |
| An8 | 4 | <u> </u> | 2 | = | 2 |
| An12 | 4 | <u> </u> | 3 | = | 1 |
| An14 | 4 | <u> </u> | 1 | = | 3 |
| An15 | 4 | _ | 2 | = | 2 |
| An16 | 4 | _ | 3 | = | 1 |
| | | Sum i | ndividual item sco | ores | 23 |

Sum individual item scores

Multiply by 13 = 299

Divide by number of items answered = 23

Fatigue Subscale Score = 23

#### SDAI[Smolen, 2003]

- The Simplified Disease Activity Index (SDAI) is a composite score consisting of the sum of SJC28, TJC28, PtGA/10, PhGA/10, and CRP (mg/dl).
- This score will be calculated based on the formula:

SDAI = SJC28 + TJC28 + PtGA / 10 + PhGA / 10 + CRP

• If one of the components is missing at an individual assessment point, the SDAI value for that assessment will be set to missing.

#### CDAI[Aletaha, 2005]

- The Clinical Disease Activity Index (CDAI) is a composite score consisting of the sum of SJC28, TJC28, PtGA/10, PhGA/10.
- This score will be calculated based on the formula:

#### CDAI = SJC28 + TJC28 + PtGA / 10 + PhGA / 10

 If one of the components is missing at an individual assessment point, the CDAI value for that assessment will be set to missing.

#### Swollen and Tender/Painful Joint Count

- Four different scores will be calculated to evaluate swelling and tenderness of joints.SJC28 and TJC28 will take 28 joints into account, SJC66 and TJC68 will use 66 and 68 joints, respectively.
- The assessment for swelling is the total number of joints with a present swelling and ranges from 0 to 28 for SJC28 and 0 to 66 for SJC66.
- The assessment for tenderness is the total number of joints with a present tenderness and ranges from 0 to 28 for TJC28 and 0 to 68 for TJC68.
- The following 28 joints will be taken into account for TJC28 and SJC28.
  - Shoulder (2 joints)
  - Knee (2)
  - Elbow (2)
  - Wrist (2)
  - Fingers (PIP, MCP: 20)
- Additionally the following joints will be taken into account for TJC68 and SJC66.
  - Temporomandibular (2)
  - Stemoclavicular (2)
  - Acromioclavicular (2)
  - Fingers (DIP: 8)
  - Ankle (2)
  - Tarsus (2)
  - o Toes (PIP, MTP: 20)
  - Hip (2, only for TJC)
- If there are missing observations for tender or swollen joints then the remaining observations will be assessed and weighted by dividing the number presented by number of non-missing and by multiplying by 28/66/68 for the joint count. No imputations for individual joints will be done. If a joint is not evaluable at Baseline, then that joint is set missing throughout the study.
- If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit.

#### Patient's Assessment of Arthritis Pain

- Subjects will assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) by placing a mark on the scale between "0" (no pain) and "10" (most severe pain), which corresponds to the magnitude of their current pain.
- Subjects will also assess the severity of their past week's arthritis pain using a continuous
  visual analogue scale (VAS) by placing a mark on the scale between "0" (no pain) and "100"
  (severe pain), which corresponds to the magnitude of their pain for the past week.
- The current endpoints are collected on eCRF after converted to a 100 unit.
- No imputations for missing data will be done.

#### Patient's Global Assessment of Disease Activity

- Subjects will complete a global assessment of disease activity using the patient global assessment (PtGA) item, a continuous VAS with anchors "0" (very well) to "10" (very poor).
- The current endpoints are collected on eCRF after converted to a 100 unit.
- No imputations for missing data will be done.

#### Physician's Global Assessment of Arthritis

- Physicians will complete a global assessment of disease activity using the physician global assessment item (PhGA), a continuous VAS with anchors "0" (none) to "10" (extremely active).
- The current endpoints are collected on eCRF after converted to a 100 unit.
- No imputations for missing data will be done.

#### 11.5.5. Immunogenicity

#### **Immunogenicity**

 Samples taken after dosing with GSK3196165 that have a value at or above the cut-point will be considered treatment emergent Anti-Drug-Antibody positive.

# 11.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

## 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as subjects who have completed all phases of the study including the following-up visit. |
| | Withdrawn subjects were not replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

# 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Binary variable | Subjects with missing efficacy data or early withdrawal will be imputed as a failure (e.g. no DAS28(CRP) remission or no moderate/good EULAR response). |
| Continuous variable | No imputation will be done. |

# 11.6.2.1. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Medications | <ul> <li>Missing start day, but month and year present: <ul> <li>If first study medication administration had been taken place in the same month and year as the occurrence of the medication, then the start day of the medication is assigned to the day of first study medication administration.</li> <li>Otherwise the start day is set to the first day of the month (eg, XX-Sep-2010 is considered as 01-Sep-2010).</li> </ul> </li> <li>Missing start day and month, but year present: <ul> <li>If first study medication administration had been taken in the same year as the occurrence of the medication, then the start date of the medication is assigned to the date of first study medication administration.</li> <li>Otherwise the start day and month is set to 01 January (eg, XX-XXX-2010 is considered as 01-Jan-2010).</li> </ul> </li> </ul> |
| | <ul> <li>Missing stop day, but month and year present:</li> <li>The day is set to the last day of the month (eg, XX-Sep-2010 is considered as 30-Sep-2010).</li> <li>Missing stop day and month, but year present:</li> <li>The stop day and month is set to 31 December (eg, XX-XXX-2010 is considered as 31-Dec-2010).</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| RA<br>diagnosis<br>and<br>symptom<br>onset | <ul> <li>Missing day, but month and year present:</li> <li>Date is set to the first day of the month.</li> <li>Missing day and month, but year present:</li> <li>Date is set to 01 January.</li> </ul> |

# 11.6.2.2. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Continuous variables | The analysis will be considered on the assumption of Missing at Random (MAR) (e.g. MMRM). |

# 11.7. Appendix 7: Multiple Comparisons & Multiplicity

No multiplicity adjustment will be planned because no formal statistical hypotheses will be tested in this study.

# 11.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### 11.8.1. Statistical Analysis Assumptions

| Endpoint(s) | • | Change from baseline in DAS28(CRP), DAS28(ESR), SDAI, CDAI and FACIT-fatigue |
|---|---|---|
| Analysis | • | MMRM |

- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

| Endpoint(s) | • | Change from baseline in DAS28(CRP) at Week 12 |
|-------------|---|-----------------------------------------------|
| Analysis | • | Dose response analysis |

 Distributional assumptions underlying the model used for analysis will be examined by obtaining a plot of the residuals versus the fitted values to gain confidence that the model assumptions are reasonable.

# 11.9. Appendix 9 – Abbreviations & Trade Marks

## 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| LOCF | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

# 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

# Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin

# 11.10. Appendix 10: List of Data Displays

# 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|-------------|
| Study Population | 1.1 to 1.21 | |
| Efficacy | 2.1 to 2.37 | 2.1 to 2.26 |
| Safety | 3.1 to 3.38 | |
| Pharmacokinetic | 4.1 to 4.4 | 4.1 to 4.8 |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.4 | 5.1 to 5.8 |
| Pharmacokinetic / Pharmacodynamic | | 6.1 to 6.3 |
| Section | List | ings |
| ICH Listings | 1 to | 77 |

# 11.10.2. Deliverable

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 11.10.3. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | | | | |
| 1.1. | ITT | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.2. | ITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC |
| 1.3. | All<br>Screening | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC |
| 1.4. | All<br>Screening | NS1 | Summary of Subjects Enrolled by Site ID | | SAC |
| Protoco | ol Deviations | | | | |
| 1.5. | Randomised | DV1 | Summary of Important Protocol Deviations | | SAC |
| Populat | Population Analysed | | | | |
| 1.6. | All<br>Screening | SP1 | Summary of Study Populations | | SAC |
| 1.7. | Randomised | SP2A | Summary of Exclusions from ITT Population | | SAC |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.8. | ITT | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.9. | ITT | POP_T5 | Summary of Baseline Efficacy Parameters | | SAC |
| 1.10. | ITT | POP_T6 | Summary of Rheumatoid factor and Anti-Cyclic Citrullinated Protein Antibody | | SAC |
| 1.11. | All<br>Screening | DM11 | Summary of Age Ranges | | SAC |
| 1.12. | ITT | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.13. | ITT | POP_T1 | Summary of Substance Use | | SAC |
| 1.14. | ITT | POP_T2 | Summary of Rheumatoid Arthritis Disease History | | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 1.15. | ITT | CM1 | Summary of Medications | | SAC |
| 1.16. | ITT | CM1 | Summary of Medications for Rheumatoid Arthritis prior to the Date of first dose | | SAC |
| 1.17. | ITT | CM1 | Summary of Medications for Rheumatoid Arthritis from the Date of first dose | | SAC |
| 1.18. | ITT | POP_T3 | Summary of Oral Corticosteroid by Visit | | SAC |
| 1.19. | ITT | POP_T3 | Summary of Change from Baseline in Oral Corticosteroid by Visit | | SAC |
| Exposi | ıre | | | | |
| 1.20. | ITT | EX1 | Summary of Exposure to Study Treatment | | SAC |
| 1.21. | ITT | POP_T4 | Summary of Exposure to MTX | | SAC |

# 11.10.4. Efficacy Tables

| Second | Secondary Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS28( | DAS28(CRP) | | | | |
| 2.1. | ITT | EFF_T1 | Summary of DAS28(CRP) Values | | SAC |
| 2.2. | ITT | EFF_T1 | Summary of Change from Baseline in DAS28(CRP) | | SAC |
| Statistic | cal Analysis fo | r DAS28(CRP) Cor | mparison with Placebo | | |
| 2.3. | ITT | EFF_T2 | Summary of Repeated Measures Analysis of Change from Baseline in DAS28(CRP) | | SAC |
| Dose R | Dose Response Analysis in DAS28(CRP) | | | | |
| 2.4. | ITT | EFF_T3 or<br>EFF_T4 | Summary of Results of Dose Response Analysis for Change from Baseline in DAS28(CRP) at Week 12 | Statistician will select the final model among the three dose response models. | SAC |

| Explora | atory Efficacy: | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| ACR 20 | /50/70 respons | ie | | | • |
| 2.5. | ITT | EFF_T5 | Summary of ACR 20 Responses | | SAC |
| 2.6. | ITT | EFF_T5 | Summary of ACR 50 Responses | | SAC |
| 2.7. | ITT | EFF_T5 | Summary of ACR 70 Responses | | SAC |
| DAS28 | (ESR) | | | | |
| 2.8. | ITT | EFF_T1 | Summary of DAS28(ESR) Values | | SAC |
| 2.9. | ITT | EFF_T1 | Summary of Change from Baseline in DAS28(ESR) | | SAC |
| 2.10. | ITT | EFF_T2 | Summary of Repeated Measures Analysis of Change from Baseline in DAS28(ESR) | | SAC |
| SDAI, C | DAI and FACIT | Γ-Fatigue | | <u> </u> | <u> </u> |
| 2.11. | ITT | EFF_T1 | Summary of SDAI Values | | SAC |
| 2.12. | ITT | EFF_T1 | Summary of CDAI Values | | SAC |
| 2.13. | ITT | EFF_T1 | Summary of FACIT-Fatigue | | SAC |
| 2.14. | ITT | EFF_T1 | Summary of Change from Baseline in SDAI | | SAC |
| 2.15. | ITT | EFF_T1 | Summary of Change from Baseline in CDAI | | SAC |
| 2.16. | ITT | EFF_T1 | Summary of Change from Baseline in FACIT-Fatigue | | SAC |
| 2.17. | ITT | EFF_T2 | Summary of Repeated Measures Analysis of Change from Baseline in SDAI | | SAC |
| 2.18. | ITT | EFF_T2 | Summary of Repeated Measures Analysis of Change from Baseline in CDAI | | SAC |
| 2.19. | ITT | EFF_T2 | Summary of Repeated Measures Analysis of Change from Baseline in FACIT-Fatigue | | SAC |

| Catego | rical DAS28(CF | RP) / DAS28(ESR) | ) Response | |
|---|---|---|---|---|
| 2.20. | ITT | EFF_T5 | Summary of Categorical DAS28(CRP) Responses | SAC |
| 2.21. | ITT | EFF_T5 | Summary of Categorical DAS28(ESR) Responses | SAC |
| DAS28 | (CRP) / DAS28( | ESR) Remission | | |
| 2.22. | ITT | EFF_T5 | Summary of DAS28(CRP) Remission | SAC |
| 2.23. | ITT | EFF_T5 | Summary of DAS28(ESR) Remission | SAC |
| The oth | ner endpoints | | | |
| 2.24. | ITT | EFF_T6 | Summary of Swollen/Tender Joint Counts | SAC |
| 2.25. | ITT | EFF_T6 | Summary of Patient's Assessment of Arthritis Pain | SAC |
| 2.26. | ITT | EFF_T1 | Summary of Patient's Global Assessment of Arthritis | SAC |
| 2.27. | ITT | EFF_T1 | Summary of Physician's Global Assessment of Arthritis | SAC |
| 2.28. | ITT | EFF_T1 | Summary of CRP | SAC |
| 2.29. | ITT | EFF_T1 | Summary of ESR | SAC |
| 2.30. | ITT | EFF_T1 | Summary of HAQ-DI score | SAC |
| 2.31. | ITT | EFF_T6 | Summary of Change from Baseline in Swollen/Tender Joint Counts | SAC |
| 2.32. | ITT | EFF_T6 | Summary of Change from Baseline in Patient's Assessment of Arthritis Pain | SAC |
| 2.33. | ITT | EFF_T1 | Summary of Change from Baseline in Patient's Global Assessment of Arthritis | SAC |
| 2.34. | ITT | EFF_T1 | Summary of Change from Baseline in Physician's Global Assessment of Arthritis | SAC |
| 2.35. | ITT | EFF_T1 | Summary of Change from Baseline in CRP | SAC |
| 2.36. | ITT | EFF_T1 | Summary of Change from Baseline in ESR | SAC |
| 2.37. | ITT | EFF_T1 | Summary of Change from Baseline in HAQ-DI score | SAC |

# 11.10.5. Efficacy Figures

| Secon | Secondary Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS28 | (CRP) | | | | |
| 2.1. | ITT | EFF_F3 | Plot of Mean (95%CI) Change from Baseline in DAS28(CRP) Profiles | | SAC |
| 2.2. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in DAS28(CRP) Profiles | | SAC |
| Statisti | cal Analysis fo | r DAS28(CRP) Co | mparison with Placebo | | |
| 2.3. | ITT | EFF_F3 | Plot of Predicted (95%CI) Treatment Difference from Placebo in DAS28(CRP) | | SAC |
| Dose R | esponse Analy | sis in DAS28(CRF | 2) | | |
| 2.4. | ITT | EFF_F2 | Plot of Predicted (95%CI) Change from Baseline in DAS28(CRP) by the final Dose Response Model at Week 12 | Statistician will select the final model among the three dose response models. | SAC |
| 2.5. | ITT | EFF_F1 | Plot of the Residuals versus the Predicted DAS28(CRP) by final Dose Response Model at Week 12 | | SAC |

| Explor | Exploratory Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| ACR20 | /50/70 | | | | • |
| 2.6. | ITT | EFF_F4 | Barplot of ACR20 Response Rate by Visit | | SAC |
| 2.7. | ITT | EFF_F4 | Barplot of ACR50 Response Rate by Visit | | SAC |
| 2.8. | ITT | EFF_F4 | Barplot of ACR70 Response Rate by Visit | | SAC |
| DAS28 | (ESR) | | | | |
| 2.9. | ITT | EFF_F3 | Plot of Mean (95%CI) Change from Baseline in DAS28(ESR) Profiles | | SAC |
| 2.10. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in DAS28(ESR) Profiles | | SAC |
| Statisti | cal Analysis fo | r DAS28(CRP) Co | mparison with Placebo | <u></u> | |
| 2.11. | ITT | EFF_F3 | Plot of Predicted (95%CI) Treatment Difference from Placebo in DAS28(ESR) | | SAC |
| SDAI, C | DAI and FACIT | -Fatigue | | | • |
| 2.12. | ITT | EFF_F3 | Plot of Mean (95%CI) Change from Baseline in SDAI Profiles | | SAC |
| 2.13. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in SDAI Profiles | | SAC |
| 2.14. | ITT | EFF_F3 | Plot of Mean (95%CI) Change from Baseline in CDAI Profiles | | SAC |
| 2.15. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in CDAI Profiles | | SAC |
| 2.16. | ITT | EFF_F3 | Plot of Mean (95%CI) Change from Baseline in FACIT-Fatigue Profiles | | SAC |
| 2.17. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in FACIT-Fatigue Profiles | | SAC |

| Explor | Exploratory Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Statisti | cal Analyses fo | or SDAI, CDAI and | FACIT-Fatigue Comparisons with Placebo | | |
| 2.18. | ITT | EFF_F3 | Plot of Predicted (95%CI) Treatment Difference from Placebo in SDAI | | SAC |
| 2.19. | ITT | EFF_F3 | Plot of Predicted (95%CI) Treatment Difference from Placebo in CDAI | | SAC |
| 2.20. | ITT | EFF_F3 | Plot of Predicted (95%CI) Treatment Difference from Placebo in FACIT-Fatigue | | SAC |
| Each C | omponents of | Composite endpo | ints | | |
| 2.21. | ITT | EFF_F3 | Plot of Mean (95% CI) Change from Baseline in CRP Profiles | | SAC |
| 2.22. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in CRP Profiles | | SAC |
| 2.23. | ITT | EFF_F3 | Plot of Mean (95% CI) Change from Baseline in ESR Profiles | | SAC |
| 2.24. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in ESR Profiles | | SAC |
| 2.25. | ITT | EFF_F3 | Plot of Mean (95% CI) Change from Baseline in HAQ-DI score Profiles | | SAC |
| 2.26. | ITT | EFF_F3 | Plot of Median (Range) Change from Baseline in HAQ-DI score Profiles | | SAC |

# 11.10.6. Safety Tables

| Safety : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Adverse Events (AEs) | | | | | |
| 3.1. | ITT | AE1 | Summary of All AEs by SOC and PT | | SAC |
| 3.2. | ITT | AE5A | Summary of All AEs by SOC and PT and Maximum Intensity | | SAC |
| 3.3. | ITT | SAFE_T4 | Summary of AESI | | SAC |
| 3.4. | ITT | AE3 | Summary of Adverse Events by Overall Frequency | | SAC |
| 3.5. | ITT | AE1 | Summary of Drug-Related AEs by SOC and PT | | SAC |
| 3.6. | ITT | AE5A | Summary of Drug-Related AEs by SOC and PT and Maximum Intensity | | SAC |
| 3.7. | ITT | AE15 | Summary of Common (>=5%) Non-Serious Adverse Events by SOC and PT | | SAC |
| 3.8. | ITT | AE1 | Summary of AEs Leading to Withdrawal from Study | | SAC |
| 3.9. | ITT | AE1 | Summary of AEs Leading to Permanent Discontinuation of Study Treatment | | SAC |
| 3.10. | ITT | SAFE_T4 | Summary of AESI Leading to Permanent Discontinuation of Study Treatment | | SAC |
| 3.11. | ITT | AE1 | Summary of Disease Related Events | | SAC |
| Serious Adverse Events (SAEs) | | | | | |
| 3.12. | ITT | AE16 | Summary of Serious Adverse Events by SOC and PT | | SAC |
| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| ECG | | | | | • |
| 3.13. | ITT | EG1 | Summary of ECG Findings | | SAC |
| 3.14. | ITT | EG2 | Summary of Change from Baseline in ECG Values by Visit | | SAC |
| 3.15. | ITT | EG2 | Summary of ECG values by visit | | SAC |
| Vital Si | gns | | | | · |
| 3.16. | ITT | VS1 | Summary of Change from Baseline in Vital Signs by Visit | | SAC |
| 3.17. | ITT | VS1 | Summary of Vital Signs by Visit | | SAC |
| Pulmor | nary | | | | · |
| 3.18. | ITT | SAFE_T1 | Summary of Cough by Visit and Grade | | SAC |
| 3.19. | ITT | SAFE_T1 | Summary of Lung Auscultation by Visit | | SAC |
| 3.20. | ITT | SAFE_T2 | Summary of Pulse Oximetry by Visit | | SAC |
| 3.21. | ITT | SAFE_T1 | Summary of Borg Dyspnea Scale by Visit | | SAC |
| 3.22. | ITT | SAFE_T2 | Summary of Percent Predicted Normal FEV1 by Visit | | SAC |
| 3.23. | ITT | SAFE_T2 | Summary of Percent Predicted Normal FVC by Visit | | SAC |
| 3.24. | ITT | SAFE_T2 | Summary of Percent Predicted HGB Corrected DLCO by Visit | | SAC |
| 3.25. | ITT | SAFE_T2 | Summary of Change from Baseline in Pulse Oximetry by Visit | | SAC |
| 3.26. | ITT | SAFE_T2 | Summary of Change from Baseline in Percent Predicted Normal FEV1 by Visit | | SAC |
| 3.27. | ITT | SAFE_T2 | Summary of Change from Baseline in Percent Predicted Normal FVC by Visit | | SAC |
| 3.28. | ITT | SAFE_T2 | Summary of Change from Baseline in Percent Predicted HGB Corrected DLCO by Visit | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Respira | atory events | | | | |
| 3.29. | ITT | SAFE_T5 | Summary of Persistent cough, dyspnea and DLCO decrease by > 15% | | SAC |
| Chemis | stry | | | | |
| 3.30. | ITT | LB1 | Summary of Chemistry Changes from Baseline | | SAC |
| 3.31. | ITT | LB1 | Summary of Chemistry by visit | | SAC |
| 3.32. | ITT | LB15 | Summary of Emergent Chemistry Results Relative to Normal Ranges | | SAC |
| Hemato | ology | | | | |
| 3.33. | ITT | LB1 | Summary of Hematology Changes from Baseline | | SAC |
| 3.34. | ITT | LB1 | Summary of Hematology by Visit | | SAC |
| 3.35. | ITT | LB15 | Summary of Emergent Hematology Results Relative to Normal Range | | SAC |
| Urinaly | sis | | | | |
| 3.36. | ITT | UR3 | Summary of Urinalysis Dipstick Results | | SAC |
| Hepato | biliary (Liver) | | | | |
| 3.37. | ITT | LIVER10 | Summary of Hepatobiliary Laboratory Abnomalities | | SAC |
| lmmun | ogenicity | | | | |
| 3.38. | Immunogeni<br>city | SAFE_T3 | Summary of Immunogenicity | | SAC |

#### 11.10.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Serum | GSK3196165 C | oncentrations | | | |
| 4.1. | PK | PK01 | Summary of Serum GSK3196165 Concentrations | | SAC |
| PK Para | ameters | | | | |
| 4.2. | PK | PK03 | Summary of Derived Serum GSK3196165 Pharmacokinetic Parameters | | SAC |
| 4.3. | PK | PK05 | Summary of Log-Transformed Derived Serum GSK3196165 Pharmacokinetic Parameters | | SAC |
| 4.4. | PK | PK_T1 | Summary of Power Model Analysis for Dose Proportionality of GSK3196165 Pharmacokinetic Parameters | <ul> <li>Cmax</li> <li>AUCtau</li> <li>AUC(0-t)</li> <li>AUC(0-inf)</li> </ul> | SAC |

# 11.10.8. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Serum | Serum GSK3196165 Concentrations | | | | |
| 4.1. | PK | PK_F1 | Individual Serum GSK3196165 Concentration-Time Plots (Linear and Semi-log) | | SAC |
| 4.2. | PK | PK17 | Mean Serum GSK3196165 Concentration-Time Plots (Linear and Semi-log) | | SAC |
| 4.3. | PK | PK18 | Median Serum GSK3196165 Concentration-Time Plots (Linear and Semi-log) | | SAC |
| Parame | eters | | | | |
| 4.4. | PK | PK28 | Plot of Individual Serum GSK3196196 Pharmacokinetic Parameters versus Dose | <ul> <li>Cmax</li> <li>AUCtau</li> <li>AUC(0-t)</li> <li>AUC(0-inf)</li> </ul> | SAC |
| 4.5. | PK | PK_F2 | Plot of GSK3196165 Pharmacokinetic Parameter Cmax vs. Treatment | | SAC |
| 4.6. | PK | PK_F2 | Plot of GSK3196165 Pharmacokinetic Parameter AUCtau vs. Treatment | | SAC |
| 4.7. | PK | PK_F2 | Plot of GSK3196165 Pharmacokinetic Parameter AUC(0-t) vs. Treatment | | SAC |
| 4.8. | PK | PK_F2 | Plot of GSK3196165 Pharmacokinetic Parameter AUC(0-inf) vs. Treatment | | SAC |

### 11.10.9. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Biomar | kers | | | · | |
| 5.1. | ITT | PD1 | Summary of Biomarkers | <ul> <li>free soluble GM-CSF</li> <li>soluble GM-CSF complexed to GSK3196165</li> <li>MRP8/14</li> <li>ARGS neopitope</li> <li>YKL-40</li> <li>14-3-3η</li> <li>IL-6</li> <li>IL-1β</li> <li>TNFα</li> <li>IL-17A</li> <li>IL-17F</li> </ul> | SAC |
| 5.2. | ITT | PD3 | Summary of Change from Baseline in Biomarkers | <ul> <li>free soluble GM-CSF</li> <li>soluble GM-CSF complexed to GSK3196165</li> <li>MRP8/14</li> <li>ARGS neopitope</li> <li>YKL-40</li> <li>14-3-3η</li> <li>IL-6</li> <li>IL-1β</li> <li>TNFα</li> <li>IL-17A</li> <li>IL-17F</li> </ul> | SAC |

| Pharmacodynamic and Biomarker : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Safety I | Biomarkers | | | | |
| 5.3. | ITT | PD1 | Summary of Safety Biomakers | <ul> <li>SP-D</li> <li>KL-6</li> <li>Cholestenoic Acid</li> <li>GM-CSF Autoantibodies at<br/>Baseline</li> </ul> | SAC |
| 5.4. | ITT | PD3 | Summary of Change from Baseline in Safety Biomarkers | <ul><li>SP-D</li><li>KL-6</li><li>Cholestenoic Acid</li></ul> | SAC |

### 11.10.10. Pharmacodynamic and Biomarker Figures

| Pharma | Pharmacodynamic and Biomarker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Biomar | kers | | | | |
| 5.1. | ITT | PD_F1 | Plot of Mean Biomarkers | <ul> <li>free soluble GM-CSF</li> <li>soluble GM-CSF complexed to GSK3196165</li> <li>MRP8/14</li> <li>ARGS neopitope</li> <li>YKL-40</li> <li>14-3-3η</li> <li>IL-6</li> <li>IL-1β</li> <li>TNFα</li> <li>IL-17A</li> <li>IL-17F</li> </ul> | SAC |
| 5.2. | ITT | PD_F2 | Plot of Median Biomarkers | <ul> <li>free soluble GM-CSF</li> <li>soluble GM-CSF complexed to GSK3196165</li> <li>MRP8/14</li> <li>ARGS neopitope</li> <li>YKL-40</li> <li>14-3-3η</li> <li>IL-6</li> <li>IL-1β</li> <li>TNFα</li> <li>IL-17A</li> <li>IL-17F</li> </ul> | SAC |

| Pharma | Pharmacodynamic and Biomarker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 5.3. | ITT | PD_F1 | Plot of Mean Change from Baseline in Biomarkers -Time Profile | <ul> <li>free soluble GM-CSF</li> <li>soluble GM-CSF complexed to GSK3196165</li> <li>MRP8/14</li> <li>ARGS neopitope</li> <li>YKL-40</li> <li>14-3-3η</li> <li>IL-6</li> <li>IL-1β</li> <li>TNFα</li> <li>IL-17A</li> <li>IL-17F</li> </ul> | SAC |
| 5.4. | ITT | PD_F2 | Plot of Median Change from Baseline in Biomarkers -Time Profile | <ul> <li>free soluble GM-CSF</li> <li>soluble GM-CSF complexed to GSK3196165</li> <li>MRP8/14</li> <li>ARGS neopitope</li> <li>YKL-40</li> <li>14-3-3η</li> <li>IL-6</li> <li>IL-1β</li> <li>TNFα</li> <li>IL-17A</li> <li>IL-17F</li> </ul> | SAC |

| Pharma | Pharmacodynamic and Biomarker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Safety | Biomarkers | | | | |
| 5.5. | ITT | PD_F1 | Plot of Mean Safety Biomarkers -Time Profile | SP-D KL-6 Cholestenoic acid | SAC |
| 5.6. | ITT | PD_F2 | Plot of Median Safety Biomarkers -Time Profile | <ul><li>SP-D</li><li>KL-6</li><li>Cholestenoic acid</li></ul> | SAC |
| 5.7. | ITT | PD_F1 | Plot of Mean Change from Baseline in Safety Biomarkers -Time Profile | <ul><li>SP-D</li><li>KL-6</li><li>Cholestenoic acid</li></ul> | SAC |
| 5.8. | ITT | PD_F2 | Plot of Median Change from Baseline in Safety Biomarkers - Time Profile | <ul><li>SP-D</li><li>KL-6</li><li>Cholestenoic acid</li></ul> | SAC |

### 11.10.11. Pharmacokinetic / Pharmacodynamic Figures

| Pharma | Pharmacokinetic / Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.1. | PK | PKPD_F1 | Linear scatter plot of Change from Baseline in freesoluble GM-CSF level at each visit versus GSK3196165 concentration values at corresponding visit | | SAC |
| 6.2. | PK | PKPD_F1 | Linear scatter plot of Change from Baseline in CRP levels at each visit versus GSK3196165 concentration values at corresponding visit | | SAC |
| 6.3. | PK | PKPD_F1 | Linear scatter plot of Change from Baseline in DAS28(CRP) measures at each visit versus GSK3196165 concentration values at corresponding visit | | SAC |

### 11.10.12. ICH Listings

| ICH : Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1. | ITT | ES2 | Listing of Reasons for Subject Withdrawal | | SAC |
| 2. | ITT | SD2 | Listing of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC |
| 3. | ALL<br>Screening | ES7 | Listing of Screening Status and Reasons for Screen Failure | | SAC |
| 4. | ALL<br>Screening | ES9 | Listing of Subjects Who Were Rescreened | | SAC |
| 5. | Randomised | BL1 | Listing of Subjects Whom the Treatment Blind was Broken | | SAC |
| 6. | ITT | TA1 | Listing of Planned and Actual Treatments | Sort by site id | SAC |
| Protoc | ol Deviations | | | | |
| 7. | All<br>Screening | DV2 | Listing of Important Protocol Deviations | | SAC |
| 8. | All<br>Screening | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tions Analysed | | | | |
| 9. | ITT | SP3 | Listing of Subjects Excluded from Any Population | | SAC |
| Demog | raphic and Bas | eline Characteris | tics | , | • |
| 10. | ITT | DM2 | Listing of Demographic Characteristics | | SAC |
| 11. | ITT | POP_L4 | Listing of Rheumatoid factor and Anti-Cyclic Citrullinated Protein Antibody | | SAC |
| 12. | ITT | DM9 | Listing of Race and Racial Combinations | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 13. | ITT | POP_L1 | Listing of Substance Use | | SAC |
| 14. | ITT | POP_L2 | Listing of Rheumatoid Arthritis Disease History | | SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 15. | ITT | MH2 | Listing of Medical Conditions | | SAC |
| 16. | ITT | CM3 | Listing of Medications | | SAC |
| 17. | ITT | CM6 | Listing of Relationship of Medication Class, Dictionary Term and Verbatim Text | | SAC |
| 18. | ITT | SP1 | Listing of Non-drug therapy | | SAC |
| Exposu | Exposure and Treatment Compliance | | | | |
| 19. | ITT | POP_L3 | Listing of Exposure to Study Treatment | | SAC |
| 20. | ITT | EX3 | Listing of Exposure to MTX | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events | | | | |
| 21. | ITT | AE8 | Listing of All Adverse Events | Including the flag of whether each AE is related to GSK3196165/Placebo and/or Methotrexate | SAC |
| 22. | ITT | SAFE_L1 | Listing of Adverse Events of Special Interest – Serious Infections, and Non Serious Pulmonary or Opportunistic Infections | | SAC |
| 23. | ITT | SAFE_L1 | Listing of Adverse Events of Special Interest – Systemic Hypersensitivity Reactions | | SAC |
| 24. | ITT | SAFE_L1 | Listing of Adverse Events of Special Interest – Injection Site Reaction | | SAC |
| 25. | ITT | AE7 | Listing of Subject Numbers for Individual AEs | | SAC |
| 26. | ITT | AE2 | Listing of Relationship Between AE SOCs, PT and Verbatim Text | | SAC |
| 27. | ITT | AE8 | Listing of Disease Related Events | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Serious | AE | | | | |
| 28. | ITT | AE8 | Listing of Serious Adverse Events | | SAC |
| ECG | | | | | |
| 29. | ITT | CP_EG3 | Listing of ECG values by Visit | | SAC |
| 30. | ITT | CP_EG5 | Listing of Abnormal ECG Findings | | SAC |
| Vital Si | gns | | | | |
| 31. | ITT | CP_VS4 | Listing of Vital Signs by Visit | | SAC |
| Pulmor | nary | | | | |
| 32. | ITT | SAFE_L2 | Listing of Cough by Visit and Grade | | SAC |
| 33. | ITT | SAFE_L2 | Listing of Lung Auscultation by Visit | | SAC |
| 34. | ITT | SAFE_L2 | Listing of Pulse Oximetry by Visit | | SAC |
| 35. | ITT | SAFE_L2 | Listing of Borg Dyspnea Scale by Visit | | SAC |
| 36. | ITT | SAFE_L2 | Listing of Percent Predicted Normal FEV1 by Visit | | SAC |
| 37. | ITT | SAFE_L2 | Listing of Percent Predicted Normal FVC by Visit | | SAC |
| 38. | ITT | SAFE_L2 | Listing of Percent Predicted HGB Corrected DLCO by Visit | | SAC |
| Respira | Respiratory events | | | | |
| 39. | ITT | SAFE_L5 | Listing of Persistent cough, dyspnea and DLCO decrease by > 15% | | SAC |
| Hepatio | B Virus | | | | |
| 40. | ITT | SAFE_L3 | Listing of HBV DNA monitoring | | SAC |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Chemis | Chemistry | | | | |
| 41. | ITT | LB5 | Listing of Chemistry by Visit | | SAC |
| Hemato | ology | | | | |
| 42. | ITT | LB5 | Listing of Hematology by Visit | | SAC |
| Urinaly | sis | | | | |
| 43. | ITT | UR2a | listing of Emergent Urinalysis Dipstick Results | | SAC |
| Immun | ogenicity | | | | |
| 44. | Immunogeni<br>city | SAFE_L4 | Listing of Immunogenicity | | SAC |
| DAS28 | | | | | |
| 45. | ITT | EFF_L1 | Listing of DAS28 Values | Including changes from baseline | SAC |
| ACR20/ | 50/70 | | | | |
| 46. | ITT | EFF_L2 | Listing of ACR20/50/70 | Including ACR components | SAC |
| Catego | rical DAS28 res | sponse / DAS28 re | mission | | |
| 47. | ITT | EFF_L3 | Listing of Categorical DAS28 response | | SAC |
| 48. | ITT | EFF_L4 | Listing of DAS28 remission | | SAC |
| SDAI, CDAI and FACIT-Fatigue | | | | | |
| 49. | ITT | EFF_L5 | Listing of SDAI Values | | SAC |
| 50. | ITT | EFF_L5 | Listing of CDAI Values | | SAC |
| 51. | ITT | EFF_L6 | Listing of FACIT-Fatigue Values | Including FACIT-fatigue components | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Other e | ndpoints | | | | |
| 52. | ITT | EFF_L7 | Listing of Swollen/Tender Joint Count | include assessment status (Y or N or ND) | SAC |
| 53. | ITT | EFF_L8 | Listing of Patient's Assessment of Arthritis Pain | | SAC |
| 54. | ITT | EFF_L9 | Listing of Patient's Global Assessment of Arthritis | | SAC |
| 55. | ITT | EFF_L9 | Listing of Physician's Global Assessment of Arthritis | | SAC |
| 56. | ITT | EFF_L10 | Listing of CRP | | SAC |
| 57. | ITT | EFF_L10 | Listing of ESR | | SAC |
| 58. | ITT | EFF_L11 | Listing of HAQ-DI score | Including HAQ-DI components | SAC |
| PK | PK | | | | |
| 59. | PK | PK07 | Listing of serum GSK3196165 concentration | | SAC |
| 60. | PK | PK_L1 | Listing of GSK3196165 Pharmacokinetic parameters | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Biomar | kers | | | | |
| 61. | ITT | PD10 | Listing of Biomarkers | <ul> <li>free soluble GM-CSF</li> <li>soluble GM-CSFcomplexed to GSK3196165</li> <li>MRP8/14</li> <li>ARGS neoepitope</li> <li>YKL-40</li> <li>14-3-3η</li> <li>IL-6</li> <li>IL-1□</li> <li>TNF□</li> <li>IL-17A</li> <li>IL-17F</li> </ul> | SAC |
| Safety I | Biomarkers | | | | |
| 62. | ITT | PD10 | Listing of Safety Biomarkers | <ul> <li>SP-D</li> <li>KL-6</li> <li>Cholestenoic Acid</li> <li>GM-CSF Autoantibodies</li> </ul> | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Hepato | biliary (Liver) | | | | |
| 63. | ITT | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping<br>Events | | SAC |
| 64. | ITT | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | SAC |
| 65. | ITT | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC |
| 66. | ITT | LIVER6 | Listing of Liver Stopping Event Information for RUCAM Score | | SAC |
| 67. | ITT | LIVER7 | Listing of Liver Biopsy Details | | SAC |
| 68. | ITT | LIVER8 | Listing of Liver Imaging Details | | SAC |
| 69. | ITT | JLE2 | Listing of Laboratory Tests (Antigen and Antibody) for Liver Events | | SAC |
| 70. | ITT | JLE3 | Listing of Laboratory Tests (DNA and RNA) for Liver Events | | SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Cardiov | ascular | | | | |
| 71. | ITT | EG5 | Listing of ECG Findings in Cardiovascular Events | | SAC |
| 72. | ITT | SAFE_L (CV1) | Listing of Subjects who had Cardiovascular Events | | SAC |
| 73. | ITT | SAFE_L (CV2) | Listing of Diagnostic Test for Cardiovascular Events | | SAC |
| 74. | ITT | SAFE_L<br>(FACV1) | Listing of Findings about Cardiovascular Events | | SAC |
| 75. | ITT | SAFE_L<br>(HRU1) | Listing of Healthcare Resource Utilization due to Cardiovascular Events | | SAC |
| 76. | ITT | SAFE_L<br>(NYHA1) | Listing of NYHA Functional Class for Cardiovascular Events | | SAC |
| 77. | ITT | SAFE_L<br>(DTH1) | Listing of Death in Cardiovascular Events | | SAC |

## 11.10.13. Non-ICH listings

| ICH : Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Dose R | Dose Response Analyses | | | | |
| 78. | ITT | EFF_L12 | SAS Output of Dose Response Analysis of Change from Baseline in DAS28(CRP) using Emax model with 3 parameters | | SAC |
| 79. | ITT | EFF_L12 | SAS Output of Dose Response Analysis of Change from Baseline in DAS28(CRP) using Emax model with 4 parameters | | SAC |
| 80. | ITT | EFF_L12 | SAS Output of Dose Response Analysis of Change from Baseline in DAS28(CRP) using Linear model | | SAC |